CLINICAL TRIAL: NCT04092452
Title: A PHASE 2A, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, 16-WEEK STUDY EVALUATING THE SAFETY AND EFFICACY OF PF-06650833, PF-06700841, AND PF-06826647 IN ADULTS WITH MODERATE TO SEVERE HIDRADENITIS SUPPURATIVA
Brief Title: A Study to Evaluate the Safety and Efficacy of PF-06650833, PF-06700841, and PF 06826647 in Adults With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C2501007
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Acne Inversa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide; PF-06700841; ropsacitinib

STUDY DESIGN:
Intervention Model Description: The treatment period is a parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): PF-06650833
  Interventions: Drug: PF-06650833
- Cohort 2 (Experimental): PF-6700841
  Interventions: Drug: PF-06700841
- Cohort 3 (Experimental): PF-06826647
  Interventions: Drug: PF-06826647
- Cohort placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06650833 — 400 mg QD
  Arms: Cohort 1
Drug: PF-06700841 — 45 mg QD
  Arms: Cohort 2
Drug: PF-06826647 — 400 mg QD
  Arms: Cohort 3
Drug: Placebo — placebo
  Arms: Cohort placebo

SUMMARY:
This is a study with 3 kinase inhibitors (PF 06650833, PF 06700841 and PF 06826647) in participants with moderate to severe HS. The study will have a maximum duration of approximately 26 weeks. This includes an up to 6-week Screening Period, a 16 week Dosing Period and a 4 week Follow up Period.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants, between 18-75, with a diagnosis of moderate to severe Hidradenitis Suppurativa

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) or positive HIV serology at screening,
* Infected with hepatitis B or hepatitis C viruses.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- United States (62):
  - The University Of Alabama At Birmingham, Birmingham, Alabama
  - The University of Alabama at Birmingham Hospital Outreach Lab, Birmingham, Alabama
  - The University of Alabama at Birmingham Investigation Drug Services Pharmacy, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Pacific Clinical Trials, Long Beach, California
  - Keck School of Medicine of University of Southern California, Los Angeles, California
  - UCSF Dermatology Clinic, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - UCSF Psoriasis and Skin Treatment Center, San Francisco, California
  - Clinical Science Institute, Santa Monica, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Dermatology Physicians of Connecticut, Shelton, Connecticut
  - Total Dermatology Care Center, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Olympian Clinical Research Largo Office, Largo, Florida
  - University of Miami Hospital, Miami, Florida
  - Tory Sullivan MD PA, North Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - MidState Skin Institute, Ocala, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - MedaPhase Inc., Newnan, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Georgia Skin Cancer and Aesthetic Dermatology, Watkinsville, Georgia
  - NorthShore University HealthSystem Dermatology Clinic, Skokie, Illinois
  - Ds Research, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Boston University General Clinical Research Unit, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University / Integrative Biosciences Center, Detroit, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Clinical Research Unit, Minneapolis, Minnesota
  - Lillihei Clinical Research Unit, Minneapolis, Minnesota
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Saint Louis University - Department of Dermatology, St Louis, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - J Woodson Clinical Studies Group, Henderson, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Health Radiology - University Physician Center, Hershey, Pennsylvania
  - Paddington Testing Company, Inc, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Dermatology and Skin Cancer Consultants, Humboldt, Tennessee
  - Clinical Research Solutions, Jackson, Tennessee
  - Dermatology and Skin Cancer Consultants, Jackson, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - University of Utah MidValley Dermatology, Murray, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Bellevue Dermatology Clinical Research Center, Bellevue, Washington
  - Bellevue Dermatology Clinic, Bellevue, Washington
  - Dermatology Associates of Seattle, Seattle, Washington
- Australia (6):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
- Canada (8):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Manna Research (London), London, Ontario
  - DermEffects, London, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de Recherche Saint-Louis, Québec
  - Alpha Recherche Clinique, Québec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kimball AB, Peeva E, Forman S, Moiin A, Khattri S, Porter ML, Mangold AR, Ghosh P, Banfield C, Oemar B. Brepocitinib, Zimlovisertib, and Ropsacitinib in Hidradenitis Suppurativa. NEJM Evid. 2024 Mar;3(3):EVIDoa2300155. doi: 10.1056/EVIDoa2300155. Epub 2024 Feb 9. PMID 38335032
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized at 60 sites in 3 countries, including Australia (N=6), United States (N=46) and Canada (N=8). A total of 194 participants (67% moderate and 33% severe hidradenitis suppurativa) were screened successfully and were randomized to 4 treatment groups.
Groups:
- Placebo: Participants were randomly assigned to receive matching placebo in a 1/3 ratio of PF-06650833 or PF-06700841 or PF-06826647.
- PF-06650833 400mg QD: PF-06650833 400mg was administered orally once daily (QD) by tablet.
- PF-06700841 45mg QD: PF-06700841 45mg was administered orally once daily (QD) by tablet.
- PF-06826647 400mg QD: PF-06826647 400mg was administered orally once daily (QD) by tablet.
Period: Overall Study
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Started | 48 | 47 | 52 | 47
Completed ((treatment completed)) | 35 | 30 | 37 | 31
Not Completed | 13 | 17 | 15 | 16
Not completed — Adverse Event | 1 | 3 | 3 | 7
Not completed — Lack of Efficacy | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 4 | 3 | 5 | 1
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 10 | 3 | 5
Not completed — Other | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD | Total
Number analyzed (Participants) | 48 | 47 | 52 | 47 | 194
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (8.95) | 39.9 (12.66) | 38.0 (11.76) | 36.6 (10.72) | 37.9 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 40 | 35 | 151
  Male | 6 | 13 | 12 | 12 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 7 | 8 | 35
  Not Hispanic or Latino | 41 | 34 | 43 | 38 | 156
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 26 | 26 | 28 | 112
  Black | 13 | 18 | 24 | 14 | 69
  Asian | 2 | 0 | 1 | 3 | 6
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Multiracial (Asian, White) | 0 | 0 | 0 | 1 | 1
  Not reported | 0 | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16- Minimum Risk (MR) [Full Analysis Set (FAS), Non-responder Imputation (NRI)].
Description: HiSCR response was defined as at least a 50% reduction in total abscess and inflammatory nodule (AN) count relative to baseline, and no increase in abscess count, and no increase in draining fistula count. Confidence interval (CI) was calculated using Blyth-Still-Casella method.
Time Frame: At week 16
Population: All participants randomized and received at least one dose of study intervention. One participant in the PF-06826647 group with missing data due to COVID-19 was excluded from the main analysis.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 46
Percentage of participants | 33.3 [22.2 to 45.5] | 34.0 [22.7 to 46.5] | 51.9 [39.7 to 64.0] | 37.0 [25.5 to 50.0]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; The null hypothesis for primary efficacy analysis was that the percentage of participants achieving HiSCR response at Week 16 was the same for the active treatment (PF-06650833, PF-06700841 or PF-06826647) and placebo. The treatment was considered superior to control if the difference was statistically significant at the overall 1-sided 0.1 level; Test type: Superiority; p = 0.4696, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 0.7, 90% CI 2-sided [-15.2 to 16.7], Standard Error of Mean 9.69
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0298, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 18.7, 90% CI 2-sided [2.7 to 34.6], Standard Error of Mean 9.71
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3606, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 3.5, 90% CI 2-sided [-12.6 to 19.6], Standard Error of Mean 9.79

2. Secondary Outcome: Percentage of Participants Achieving HiSCR Response at Weeks 1, 2, 4, 6, 8, and 12 - MR (FAS, NRI).
Description: as for outcome 1
Time Frame: At weeks 1, 2, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percentage of participants
  Week 1 | 16.7 [8.6 to 27.7] | 12.8 [5.7 to 22.7] | 15.4 [7.9 to 25.4] | 21.3 [12.0 to 32.2]
  Week 2: number analyzed (Participants) | 48 | 47 | 50 | 46
  Week 2 | 25.0 [15.1 to 36.9] | 31.9 [20.8 to 44.4] | 32.0 [21.2 to 43.4] | 28.3 [17.6 to 40.4]
  Week 4: number analyzed (Participants) | 47 | 47 | 51 | 47
  Week 4 | 31.9 [20.8 to 44.4] | 40.4 [28.3 to 53.5] | 39.2 [27.7 to 51.6] | 27.7 [17.2 to 40.3]
  Week 6: number analyzed (Participants) | 48 | 47 | 52 | 46
  Week 6 | 37.5 [26.4 to 50.0] | 38.3 [27.1 to 51.3] | 44.2 [32.4 to 56.3] | 41.3 [29.0 to 54.5]
  Week 8: number analyzed (Participants) | 48 | 47 | 52 | 46
  Week 8 | 43.8 [31.5 to 56.6] | 36.2 [25.1 to 48.7] | 44.2 [32.4 to 56.3] | 41.3 [29.0 to 54.5]
  Week 12: number analyzed (Participants) | 48 | 47 | 52 | 46
  Week 12 | 41.7 [29.6 to 54.5] | 31.9 [20.8 to 44.4] | 50.0 [37.9 to 62.1] | 41.3 [29.0 to 54.5]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -3.8, 90% CI 2-sided [-15.6 to 8.0], Standard Error of Mean 7.19
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -0.9, 90% CI 2-sided [-12.9 to 11.1], Standard Error of Mean 7.28
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = 4.6, 90% CI 2-sided [-8.5 to 17.8], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 7.9, 90% CI 2-sided [-6.9 to 22.8], Standard Error of Mean 9.02
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 7.5, 90% CI 2-sided [-7.1 to 22.2], Standard Error of Mean 8.91
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 3.5, 90% CI 2-sided [-11.3 to 18.3], Standard Error of Mean 9.00
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 9.0, 90% CI 2-sided [-7.1 to 25.1], Standard Error of Mean 9.79
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 7.7, 90% CI 2-sided [-8.0 to 23.5], Standard Error of Mean 9.57
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -4.0, 90% CI 2-sided [-19.4 to 11.4], Standard Error of Mean 9.37
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 0.8, 90% CI 2-sided [-15.6 to 17.2], Standard Error of Mean 9.96
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 6.7, 90% CI 2-sided [-9.4 to 22.9], Standard Error of Mean 9.81
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 3.7, 90% CI 2-sided [-12.8 to 20.2], Standard Error of Mean 10.05
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; p = 0.7798, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -7.8, 90% CI 2-sided [-24.2 to 8.7], Standard Error of Mean 9.98
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; p = 0.4819, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 0.5, 90% CI 2-sided [-15.9 to 16.8], Standard Error of Mean 9.92
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; p = 0.5933, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -2.4, 90% CI 2-sided [-19.2 to 14.4], Standard Error of Mean 10.19
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; p = 0.8421, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -9.9, 90% CI 2-sided [-26.1 to 6.2], Standard Error of Mean 9.81
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; p = 0.2090, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 8.0, 90% CI 2-sided [-8.2 to 24.2], Standard Error of Mean 9.85
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; p = 0.5183, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -0.5, 90% CI 2-sided [-17.1 to 16.2], Standard Error of Mean 10.12

3. Secondary Outcome: Percentage of Participants Achieving a Total Abscess and Inflammatory Nodule (AN) Count of 0 or 1; 0, 1 or 2 at Week 16 - MR (FAS, NRI).
Description: This estimand was intended to provide difference between treated and placebo in percentage of participants with a total AN count of 0 or 1, or 0, 1 or 2, respectively at week 16. Confidence interval (CI) was calculated using Blyth-Still-Casella method.
Time Frame: At week 16
Population: All participants randomized and received at least one dose of study intervention. In PF-06826647 400mg QD treatment group, 1 participant discontinued the study due to COVID-19 pandemic during study Days 9 - 16. Based on the pre-specification in the statistical analysis plan (SAP), this participant was excluded from the analysis after the treatment discontinuation visit.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 46
Percentage of participants
  Total AN Count of 0 or 1 | 16.7 [8.6 to 27.7] | 17.0 [8.8 to 28.3] | 28.8 [18.7 to 39.7] | 23.9 [15.1 to 35.0]
  Total AN Count of 0, 1 or 2 | 22.9 [14.4 to 34.0] | 27.7 [17.2 to 40.3] | 38.5 [27.1 to 50.0] | 32.6 [21.3 to 45.5]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Total AN Count of 0 or 1; Test type: Superiority; p = 0.5150, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -0.3, 90% CI 2-sided [-12.7 to 12.1], Standard Error of Mean 7.54
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Total AN Count of 0 or 1; Test type: Superiority; p = 0.0737, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 12.2, 90% CI 2-sided [-1.4 to 25.8], Standard Error of Mean 8.28
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Total AN Count of 0 or 1; Test type: Superiority; p = 0.2081, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 6.6, 90% CI 2-sided [-6.7 to 20.0], Standard Error of Mean 8.11
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Total AN Count of 0, 1 or 2; Test type: Superiority; p = 0.2957, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 4.8, 90% CI 2-sided [-9.9 to 19.4], Standard Error of Mean 8.90
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Total AN Count of 0, 1 or 2; Test type: Superiority; p = 0.0456, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 15.6, 90% CI 2-sided [0.7 to 30.5], Standard Error of Mean 9.07
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Total AN Count of 0, 1 or 2; Test type: Superiority; p = 0.1558, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 9.2, 90% CI 2-sided [-5.7 to 24.1], Standard Error of Mean 9.05

4. Secondary Outcome: Least Squares (LS) Mean of Percent Change From Baseline in AN Count at Weeks 1, 2, 4, 6, 8, 12 and 16 - Analysis of Covariance (ANCOVA) [FAS, Multiply Imputed (MI)].
Description: The analysis of covariance (ANCOVA) model was implemented for statistical testing, which included terms of treatment group, the stratification factors, and the baseline value as the independent variable.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percent change
  Week 1: number analyzed (Participants) | 45 | 42 | 45 | 41
  Week 1 | -1.94 [-12.37 to 8.50] | -13.92 [-24.50 to -3.35] | -17.00 [-27.35 to -6.66] | -19.39 [-30.40 to -8.38]
  Week 2: number analyzed (Participants) | 46 | 42 | 44 | 43
  Week 2 | -22.29 [-33.70 to -10.88] | -34.81 [-46.81 to -22.82] | -25.15 [-36.73 to -13.57] | -27.79 [-39.61 to -15.96]
  Week 4: number analyzed (Participants) | 45 | 42 | 42 | 34
  Week 4 | -26.46 [-40.31 to -12.61] | -30.98 [-44.77 to -17.18] | -44.00 [-57.40 to -30.59] | -30.38 [-45.18 to -15.58]
  Week 6: number analyzed (Participants) | 43 | 40 | 41 | 34
  Week 6 | -33.05 [-49.47 to -16.64] | -25.96 [-42.45 to -9.47] | -47.62 [-64.49 to -30.75] | -42.00 [-59.13 to -24.87]
  Week 8: number analyzed (Participants) | 43 | 39 | 44 | 36
  Week 8 | -36.26 [-52.53 to -19.98] | -24.76 [-40.74 to -8.77] | -52.41 [-68.05 to -36.76] | -51.33 [-68.17 to -34.48]
  Week 12: number analyzed (Participants) | 40 | 34 | 41 | 32
  Week 12 | -32.52 [-50.98 to -14.06] | -39.06 [-58.63 to -19.48] | -49.70 [-65.92 to -33.47] | -52.51 [-70.36 to -34.66]
  Week 16: number analyzed (Participants) | 35 | 29 | 37 | 30
  Week 16 | -34.96 [-59.85 to -10.07] | -24.11 [-49.42 to 1.20] | -52.58 [-76.77 to -28.39] | -44.37 [-69.80 to -18.94]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -11.98, 90% CI 2-sided [-26.16 to 2.20], Standard Error of Mean 8.622
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -15.07, 90% CI 2-sided [-29.09 to -1.04], Standard Error of Mean 8.526
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -17.45, 90% CI 2-sided [-31.86 to -3.05], Standard Error of Mean 8.758
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = -12.52, 90% CI 2-sided [-28.09 to 3.05], Standard Error of Mean 9.465
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = -2.86, 90% CI 2-sided [-18.22 to 12.50], Standard Error of Mean 9.338
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = -5.50, 90% CI 2-sided [-21.02 to 10.03], Standard Error of Mean 9.438
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -4.52, 90% CI 2-sided [-22.96 to 13.93], Standard Error of Mean 11.214
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -17.54, 90% CI 2-sided [-35.84 to 0.77], Standard Error of Mean 11.131
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -3.92, 90% CI 2-sided [-22.85 to 15.00], Standard Error of Mean 11.507
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 7.09, 90% CI 2-sided [-15.04 to 29.22], Standard Error of Mean 13.452
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = -14.57, 90% CI 2-sided [-37.08 to 7.95], Standard Error of Mean 13.688
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = -8.95, 90% CI 2-sided [-31.66 to 13.76], Standard Error of Mean 13.808
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; p = 0.8108, ANCOVA — One-sided p-value; Risk Difference (RD) = 11.50, 90% CI 2-sided [-9.98 to 32.98], Standard Error of Mean 13.057
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; p = 0.1043, ANCOVA — One-sided p-value; Risk Difference (RD) = -16.15, 90% CI 2-sided [-37.28 to 4.98], Standard Error of Mean 12.845
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; p = 0.1296, ANCOVA — One-sided p-value; Risk Difference (RD) = -15.07, 90% CI 2-sided [-37.04 to 6.90], Standard Error of Mean 13.355
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; p = 0.3450, ANCOVA — One-sided p-value; Risk Difference (RD) = -6.54, 90% CI 2-sided [-33.49 to 20.42], Standard Error of Mean 16.384
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; p = 0.1119, ANCOVA — One-sided p-value; Risk Difference (RD) = -17.18, 90% CI 2-sided [-40.40 to 6.04], Standard Error of Mean 14.116
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; p = 0.0885, ANCOVA — One-sided p-value; Risk Difference (RD) = -19.99, 90% CI 2-sided [-44.34 to 4.37], Standard Error of Mean 14.806
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; p = 0.7050, ANCOVA — One-sided p-value; Risk Difference (RD) = 10.85, 90% CI 2-sided [-22.28 to 43.98], Standard Error of Mean 20.140
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; p = 0.1833, ANCOVA — One-sided p-value; Risk Difference (RD) = -17.62, 90% CI 2-sided [-49.73 to 14.48], Standard Error of Mean 19.519
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; p = 0.3213, ANCOVA — One-sided p-value; Risk Difference (RD) = -9.41, 90% CI 2-sided [-42.76 to 23.94], Standard Error of Mean 20.277

5. Secondary Outcome: Least Squares Mean of Absolute Score in International Hidradenitis Suppurativa Severity Score System (IHS4) at Weeks 1, 2, 4, 6, 8, 12 and 16 - ANCOVA (FAS, MI).
Description: The IHS4 score was calculated by the number of nodules, the number of abscesses, and the number of draining tunnels. IHS4 score = (number of nodules × 1) + (number of abscesses × 2) + {number of draining tunnels (fistulae/sinuses) × 4}. Confidence interval (CI) was calculated using Blyth-Still-Casella method. Lower IHS4 absolute scores mean a better outcome.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Units on a scale
  Week 1 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 45 | 42 | 45 | 42
  Week 1 - Statistical Analysis (MI) - Absolute Score | 22.9 [19.6 to 26.1] | 21.4 [18.1 to 24.6] | 20.8 [17.7 to 24.0] | 21.4 [18.1 to 24.7]
  Week 2 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 2 - Statistical Analysis (MI) - Absolute Score | 18.9 [15.8 to 22.1] | 18.0 [14.8 to 21.2] | 18.8 [15.7 to 21.9] | 19.0 [15.7 to 22.2]
  Week 4 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 45 | 42 | 42 | 35
  Week 4 - Statistical Analysis (MI) - Absolute Score | 17.9 [14.8 to 20.9] | 17.5 [14.4 to 20.6] | 16.5 [13.6 to 19.5] | 13.3 [10.0 to 16.7]
  Week 6 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 43 | 40 | 41 | 35
  Week 6 - Statistical Analysis (MI) - Absolute Score | 19.7 [16.0 to 23.3] | 18.1 [14.4 to 21.7] | 14.9 [11.4 to 18.5] | 14.2 [10.3 to 18.1]
  Week 8 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 43 | 39 | 44 | 37
  Week 8 - Statistical Analysis (MI) - Absolute Score | 14.9 [11.5 to 18.3] | 15.9 [12.5 to 19.4] | 15.0 [11.7 to 18.4] | 11.1 [7.5 to 14.7]
  Week 12 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 40 | 34 | 41 | 33
  Week 12 - Statistical Analysis (MI) - Absolute Score | 15.8 [12.6 to 18.9] | 14.5 [11.2 to 17.8] | 13.0 [10.0 to 16.0] | 12.9 [9.5 to 16.3]
  Week 16 - Statistical Analysis (MI) - Absolute Score: number analyzed (Participants) | 35 | 29 | 37 | 30
  Week 16 - Statistical Analysis (MI) - Absolute Score | 16.0 [12.4 to 19.6] | 13.4 [9.5 to 17.3] | 12.0 [8.8 to 15.3] | 13.4 [9.8 to 17.0]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -1.5, 90% CI 2-sided [-5.9 to 2.9], Standard Error of Mean 2.67
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -2.0, 90% CI 2-sided [-6.3 to 2.2], Standard Error of Mean 2.60
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -1.5, 90% CI 2-sided [-5.9 to 2.9], Standard Error of Mean 2.68
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -0.9, 90% CI 2-sided [-5.2 to 3.3], Standard Error of Mean 2.59
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -0.1, 90% CI 2-sided [-4.3 to 4.1], Standard Error of Mean 2.55
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = 0.0, 90% CI 2-sided [-4.3 to 4.3], Standard Error of Mean 2.61
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -0.3, 90% CI 2-sided [-4.5 to 3.8], Standard Error of Mean 2.51
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -1.3, 90% CI 2-sided [-5.4 to 2.8], Standard Error of Mean 2.48
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -4.5, 90% CI 2-sided [-8.8 to -0.3], Standard Error of Mean 2.58
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -1.6, 90% CI 2-sided [-6.5 to 3.3], Standard Error of Mean 2.99
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -4.7, 90% CI 2-sided [-9.5 to 0.1], Standard Error of Mean 2.91
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; Risk Difference (RD) = -5.4, 90% CI 2-sided [-10.5 to -0.4], Standard Error of Mean 3.08
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.6393, ANCOVA — One-sided p-value; Risk Difference (RD) = 1.0, 90% CI 2-sided [-3.6 to 5.6], Standard Error of Mean 2.78
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.5178, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.1, 90% CI 2-sided [-4.4 to 4.6], Standard Error of Mean 2.72
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.0864, ANCOVA — One-sided p-value; Risk Difference (RD) = -3.8, 90% CI 2-sided [-8.5 to 0.8], Standard Error of Mean 2.82
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.3172, ANCOVA — One-sided p-value; Risk Difference (RD) = -1.2, 90% CI 2-sided [-5.5 to 3.1], Standard Error of Mean 2.61
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.1384, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.7, 90% CI 2-sided [-6.8 to 1.4], Standard Error of Mean 2.51
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.1427, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.8, 90% CI 2-sided [-7.2 to 1.5], Standard Error of Mean 2.66
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.1975, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.5, 90% CI 2-sided [-7.5 to 2.4], Standard Error of Mean 2.99
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.0755, ANCOVA — One-sided p-value; Risk Difference (RD) = -4.0, 90% CI 2-sided [-8.5 to 0.6], Standard Error of Mean 2.76
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 - Statistical Analysis (MI) - Absolute Score; Test type: Superiority; p = 0.1869, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.6, 90% CI 2-sided [-7.3 to 2.2], Standard Error of Mean 2.89

6. Secondary Outcome: Least Squares Mean of Percent Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) at Weeks 1, 2, 4, 6, 8, 12 and 16 - ANCOVA (FAS, MI).
Description: as for outcome 5
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percent change
  Week 1 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 45 | 42 | 45 | 42
  Week 1 - Statistical Analysis (MI) - Percent Change from Baseline | -7.26 [-17.77 to 3.26] | -10.91 [-21.57 to -0.25] | -21.02 [-31.75 to -10.30] | -24.77 [-35.94 to -13.59]
  Week 2 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 2 - Statistical Analysis (MI) - Percent Change from Baseline | -26.58 [-38.80 to -14.37] | -30.87 [-43.51 to -18.23] | -28.63 [-40.68 to -16.59] | -26.41 [-38.99 to -13.84]
  Week 4 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 45 | 42 | 42 | 35
  Week 4 - Statistical Analysis (MI) - Percent Change from Baseline | -32.64 [-45.55 to -19.72] | -33.10 [-45.56 to -20.65] | -40.71 [-52.76 to -28.66] | -38.70 [-52.26 to -25.14]
  Week 6 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 43 | 40 | 41 | 35
  Week 6 - Statistical Analysis (MI) - Percent Change from Baseline | -30.57 [-45.47 to -15.67] | -34.10 [-49.16 to -19.05] | -46.83 [-62.62 to -31.03] | -43.09 [-59.05 to -27.13]
  Week 8 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 43 | 39 | 44 | 37
  Week 8 - Statistical Analysis (MI) - Percent Change from Baseline | -41.30 [-54.94 to -27.67] | -35.51 [-49.04 to -21.98] | -47.12 [-60.38 to -33.85] | -52.64 [-67.14 to -38.14]
  Week 12 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 40 | 34 | 41 | 33
  Week 12 - Statistical Analysis (MI) - Percent Change from Baseline | -36.46 [-50.16 to -22.76] | -43.24 [-56.66 to -29.82] | -53.03 [-65.59 to -40.47] | -50.11 [-65.53 to -34.70]
  Week 16 - Statistical Analysis (MI) - Percent Change from Baseline: number analyzed (Participants) | 35 | 29 | 37 | 30
  Week 16 - Statistical Analysis (MI) - Percent Change from Baseline | -37.84 [-54.85 to -20.82] | -43.47 [-60.47 to -26.47] | -52.64 [-70.79 to -34.49] | -46.16 [-64.20 to -28.11]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -3.65, 90% CI 2-sided [-17.90 to 10.59], Standard Error of Mean 8.659
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -13.77, 90% CI 2-sided [-28.16 to 0.62], Standard Error of Mean 8.749
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -17.51, 90% CI 2-sided [-31.91 to -3.12], Standard Error of Mean 8.752
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -4.29, 90% CI 2-sided [-20.91 to 12.33], Standard Error of Mean 10.103
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -2.05, 90% CI 2-sided [-18.34 to 14.24], Standard Error of Mean 9.904
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = 0.17, 90% CI 2-sided [-16.34 to 16.68], Standard Error of Mean 10.039
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -0.46, 90% CI 2-sided [-17.29 to 16.36], Standard Error of Mean 10.227
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -8.07, 90% CI 2-sided [-24.77 to 8.63], Standard Error of Mean 10.155
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -6.06, 90% CI 2-sided [-23.35 to 11.22], Standard Error of Mean 10.509
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -3.54, 90% CI 2-sided [-23.71 to 16.63], Standard Error of Mean 12.262
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -16.26, 90% CI 2-sided [-36.84 to 4.32], Standard Error of Mean 12.510
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; Risk Difference (RD) = -12.52, 90% CI 2-sided [-33.27 to 8.22], Standard Error of Mean 12.610
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.7000, ANCOVA — One-sided p-value; Risk Difference (RD) = 5.79, 90% CI 2-sided [-12.38 to 23.96], Standard Error of Mean 11.045
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.2965, ANCOVA — One-sided p-value; Risk Difference (RD) = -5.81, 90% CI 2-sided [-23.70 to 12.08], Standard Error of Mean 10.876
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.1568, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.33, 90% CI 2-sided [-29.83 to 7.17], Standard Error of Mean 11.247
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.2672, ANCOVA — One-sided p-value; Risk Difference (RD) = -6.78, 90% CI 2-sided [-24.73 to 11.17], Standard Error of Mean 10.912
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.0576, ANCOVA — One-sided p-value; Risk Difference (RD) = -16.57, 90% CI 2-sided [-33.87 to 0.73], Standard Error of Mean 10.517
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.1197, ANCOVA — One-sided p-value; Risk Difference (RD) = -13.65, 90% CI 2-sided [-32.74 to 5.44], Standard Error of Mean 11.603
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.3388, ANCOVA — One-sided p-value; Risk Difference (RD) = -5.63, 90% CI 2-sided [-27.91 to 16.65], Standard Error of Mean 13.545
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 - Statistical Analysis (MI) - Percent Change from Baseline; Test type: Superiority; p = 0.1376, ANCOVA — One-sided p-value; Risk Difference (RD) = -14.80, 90% CI 2-sided [-37.12 to 7.51], Standard Error of Mean 13.567
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; p = 0.2741, ANCOVA — One-sided p-value; Risk Difference (RD) = -8.32, 90% CI 2-sided [-31.12 to 14.48], Standard Error of Mean 13.860

7. Secondary Outcome: Percentage of Participants Who Experienced a Hidradenitis Suppurativa (HS) Flare at Weeks 4, 8, 12 and 16 - MR [FAS, Only Observed Data (OBS)].
Description: HS flare was defined as at least a 25% increase in AN count with a minimum increase of 2 relative to Baseline. Confidence interval (CI) was calculated using Blyth-Still-Casella method.
Time Frame: At weeks 4, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percentage of participants
  Week 4: number analyzed (Participants) | 45 | 42 | 42 | 35
  Week 4 | 13.3 [6.0 to 23.7] | 11.9 [5.9 to 22.7] | 4.8 [1.3 to 13.5] | 14.3 [7.1 to 26.0]
  Week 8: number analyzed (Participants) | 43 | 39 | 44 | 37
  Week 8 | 9.3 [4.1 to 18.9] | 15.4 [6.9 to 27.7] | 2.3 [0.2 to 9.4] | 0 [0.0 to 7.3]
  Week 12: number analyzed (Participants) | 40 | 34 | 41 | 33
  Week 12 | 17.5 [9.5 to 29.2] | 5.9 [1.6 to 16.9] | 2.4 [0.3 to 10.1] | 0 [0.0 to 8.2]
  Week 16: number analyzed (Participants) | 35 | 29 | 37 | 30
  Week 16 | 17.1 [7.7 to 30.2] | 6.9 [1.8 to 20.0] | 0 [0.0 to 7.3] | 3.3 [0.4 to 14.0]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -1.3, 90% CI 2-sided [-13.0 to 10.3], Standard Error of Mean 7.06
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -8.5, 90% CI 2-sided [-18.7 to 1.8], Standard Error of Mean 6.23
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 1.7, 90% CI 2-sided [-10.7 to 14.1], Standard Error of Mean 7.55
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; p = 0.8372, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 6.6, 90% CI 2-sided [-4.6 to 17.7], Standard Error of Mean 6.80
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; p = 0.0819, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -6.4, 90% CI 2-sided [-14.1 to 1.3], Standard Error of Mean 4.68
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; p = 0.0242, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -8.0, 90% CI 2-sided [-15.2 to -0.9], Standard Error of Mean 4.34
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; p = 0.0264, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -12.7, 90% CI 2-sided [-23.1 to -2.3], Standard Error of Mean 6.33
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; p = 0.0127, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -14.5, 90% CI 2-sided [-25.1 to -3.9], Standard Error of Mean 6.47
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; p = 0.0059, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -16.6, 90% CI 2-sided [-27.0 to -6.2], Standard Error of Mean 6.33
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; p = 0.1185, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -9.6, 90% CI 2-sided [-22.7 to 3.5], Standard Error of Mean 7.97
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; p = 0.0040, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -16.1, 90% CI 2-sided [-26.6 to -5.6], Standard Error of Mean 6.39
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; p = 0.0418, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -12.8, 90% CI 2-sided [-24.5 to -1.1], Standard Error of Mean 7.09

8. Secondary Outcome: Percentage of Participants Achieving Skin Pain Numeric Rating Scale (NRS30), at Worst, at Weeks 1, 2, 4, 6, 8, 12 and 16 - MR (FAS With Baseline ≥3, NRI)
Description: The rate comparing treatment and placebo groups at each visit was analyzed using CMH test with MR weighting strategy between each of active treatment group and placebo. Confidence interval (CI) was calculated using Blyth-Still-Casella method. NRS30 was defined as ≥30% reduction and ≥1 unit reduction from baseline in Patient's Global Assessment (PGA) Skin Pain NRS. The range of skin pain was from 0 to 10. Lower IHS4 absolute scores mean a better outcome. Baseline was defined as the average of all values recorded between Day -6 and Day 1. Weekly data were average values of daily observations over 7 days. NRI (non-responder imputation) for missing values which were related to withdrawal and all other events except for COVID-19.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention with baseline NRS≥3 scores. One participant in the PF-06826647 group with missing data due to COVID-19 was excluded from the main analysis.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 41 | 37 | 42 | 41
Percentage of participants
  Week 1 (Pain at its Worst) | 7.3 [2.7 to 17.3] | 18.9 [10.4 to 31.8] | 16.7 [9.1 to 27.7] | 19.5 [10.1 to 31.2]
  Week 2 (Pain at its Worst) | 17.1 [9.3 to 28.4] | 21.6 [11.2 to 34.3] | 28.6 [17.4 to 41.0] | 24.4 [13.9 to 37.4]
  Week 4 (Pain at its Worst) | 34.1 [23.0 to 46.9] | 16.2 [7.3 to 29.3] | 40.5 [27.7 to 54.3] | 31.7 [19.9 to 44.5]
  Week 6 (Pain at its Worst) | 41.5 [28.4 to 55.5] | 21.6 [11.2 to 34.3] | 38.1 [25.6 to 52.0] | 29.3 [17.8 to 42.1]
  Week 8 (Pain at its Worst): number analyzed (Participants) | 41 | 37 | 42 | 40
  Week 8 (Pain at its Worst) | 34.1 [23.0 to 46.9] | 29.7 [18.5 to 43.3] | 50.0 [36.5 to 63.5] | 27.5 [17.5 to 40.9]
  Week 12 (Pain at its Worst): number analyzed (Participants) | 41 | 37 | 42 | 40
  Week 12 (Pain at its Worst) | 43.9 [31.2 to 57.9] | 29.7 [18.5 to 43.3] | 40.5 [27.7 to 54.3] | 35.0 [23.4 to 48.3]
  Week 16 (Pain at its Worst): number analyzed (Participants) | 41 | 37 | 42 | 40
  Week 16 (Pain at its Worst) | 29.3 [17.8 to 42.1] | 21.6 [11.2 to 34.3] | 35.7 [23.7 to 48.0] | 35.0 [23.4 to 48.3]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 (Pain at its Worst); Test type: Superiority; p = 0.0559, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 12.1, 90% CI 2-sided [-0.7 to 24.8], Standard Error of Mean 7.75
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 (Pain at its Worst); Test type: Superiority; p = 0.0758, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 9.8, 90% CI 2-sided [-1.9 to 21.4], Standard Error of Mean 7.09
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 (Pain at its Worst); Test type: Superiority; p = 0.0637, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 11.3, 90% CI 2-sided [-0.6 to 23.2], Standard Error of Mean 7.21
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 (Pain at its Worst); Test type: Superiority; p = 0.3179, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 4.2, 90% CI 2-sided [-10.3 to 18.8], Standard Error of Mean 8.84
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 (Pain at its Worst); Test type: Superiority; p = 0.1078, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 11.0, 90% CI 2-sided [-3.5 to 25.5], Standard Error of Mean 8.82
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 (Pain at its Worst); Test type: Superiority; p = 0.1976, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 7.6, 90% CI 2-sided [-7.0 to 22.2], Standard Error of Mean 8.86
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 (Pain at its Worst); Test type: Superiority; p = 0.9738, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -18.9, 90% CI 2-sided [-34.3 to -3.6], Standard Error of Mean 9.32
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 (Pain at its Worst); Test type: Superiority; p = 0.2925, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 5.8, 90% CI 2-sided [-11.3 to 22.9], Standard Error of Mean 10.40
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 (Pain at its Worst); Test type: Superiority; p = 0.6178, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -3.1, 90% CI 2-sided [-19.8 to 13.7], Standard Error of Mean 10.18
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 (Pain at its Worst); Test type: Superiority; p = 0.9769, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -20.9, 90% CI 2-sided [-37.4 to -4.4], Standard Error of Mean 10.04
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 (Pain at its Worst); Test type: Superiority; p = 0.6529, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -4.2, 90% CI 2-sided [-21.6 to 13.2], Standard Error of Mean 10.57
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 (Pain at its Worst); Test type: Superiority; p = 0.8878, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -12.8, 90% CI 2-sided [-29.8 to 4.3], Standard Error of Mean 10.36
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 (Pain at its Worst); Test type: Superiority; p = 0.7259, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -6.2, 90% CI 2-sided [-22.9 to 10.4], Standard Error of Mean 10.11
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 (Pain at its Worst); Test type: Superiority; p = 0.0826, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 14.8, 90% CI 2-sided [-2.1 to 31.6], Standard Error of Mean 10.24
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 (Pain at its Worst); Test type: Superiority; p = 0.7884, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -8.0, 90% CI 2-sided [-24.1 to 8.0], Standard Error of Mean 9.75
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 (Pain at its Worst); Test type: Superiority; p = 0.9326, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -16.1, 90% CI 2-sided [-33.2 to 1.1], Standard Error of Mean 10.43
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 (Pain at its Worst); Test type: Superiority; p = 0.6810, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -4.9, 90% CI 2-sided [-22.1 to 12.2], Standard Error of Mean 10.41
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 (Pain at its Worst); Test type: Superiority; p = 0.8308, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -10.3, 90% CI 2-sided [-27.6 to 7.0], Standard Error of Mean 10.52
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 (Pain at its Worst); Test type: Superiority; p = 0.8063, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -8.5, 90% CI 2-sided [-24.5 to 7.4], Standard Error of Mean 9.71
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 (Pain at its Worst); Test type: Superiority; p = 0.2649, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 6.5, 90% CI 2-sided [-10.4 to 23.4], Standard Error of Mean 10.27
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 (Pain at its Worst); Test type: Superiority; p = 0.3029, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 5.3, 90% CI 2-sided [-11.7 to 22.4], Standard Error of Mean 10.35

9. Secondary Outcome: Percentage of Participants Achieving Skin Pain Numeric Rating Scale (NRS30), on Average, at Weeks 1, 2, 4, 6, 8, 12 and 16 - MR (FAS With Baseline ≥3, NRI)
Description: as for outcome 8
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 39 | 34 | 41 | 35
Percentage of participants
  Week 1 (Average Pain) | 10.3 [4.5 to 21.0] | 17.6 [8.0 to 30.7] | 24.4 [13.9 to 37.4] | 8.6 [3.2 to 19.3]
  Week 2 (Average Pain) | 17.9 [9.8 to 30.0] | 20.6 [11.3 to 34.9] | 36.6 [24.6 to 50.0] | 22.9 [11.9 to 36.5]
  Week 4 (Average Pain) | 33.3 [21.0 to 47.1] | 20.6 [11.3 to 34.9] | 46.3 [33.9 to 60.2] | 34.3 [22.0 to 47.8]
  Week 6 (Average Pain) | 48.7 [35.6 to 61.9] | 32.4 [19.7 to 46.2] | 48.8 [35.1 to 62.6] | 34.3 [22.0 to 47.8]
  Week 8 (Average Pain): number analyzed (Participants) | 39 | 34 | 41 | 34
  Week 8 (Average Pain) | 35.9 [23.9 to 50.0] | 26.5 [15.9 to 40.5] | 56.1 [42.1 to 68.8] | 29.4 [16.9 to 43.3]
  Week 12 (Average Pain): number analyzed (Participants) | 39 | 34 | 41 | 34
  Week 12 (Average Pain) | 41.0 [27.7 to 55.4] | 26.5 [15.9 to 40.5] | 41.5 [28.4 to 55.5] | 32.4 [19.7 to 46.2]
  Week 16 (Average Pain): number analyzed (Participants) | 39 | 34 | 41 | 34
  Week 16 (Average Pain) | 28.2 [17.8 to 42.1] | 20.6 [11.3 to 34.9] | 39.0 [26.2 to 53.1] | 32.4 [19.7 to 46.2]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 (Average Pain); Test type: Superiority; p = 0.1687, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 7.7, 90% CI 2-sided [-5.7 to 21.2], Standard Error of Mean 8.20
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 (Average Pain); Test type: Superiority; p = 0.0376, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 13.8, 90% CI 2-sided [0.6 to 27.0], Standard Error of Mean 8.03
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 (Average Pain); Test type: Superiority; p = 0.5883, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -1.5, 90% CI 2-sided [-12.9 to 9.8], Standard Error of Mean 6.90
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 (Average Pain); Test type: Superiority; p = 0.3829, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 2.7, 90% CI 2-sided [-12.2 to 17.6], Standard Error of Mean 9.07
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 (Average Pain); Test type: Superiority; p = 0.0316, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 18.2, 90% CI 2-sided [2.5 to 33.9], Standard Error of Mean 9.54
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 (Average Pain); Test type: Superiority; p = 0.3072, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 4.6, 90% CI 2-sided [-10.5 to 19.7], Standard Error of Mean 9.17
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 (Average Pain); Test type: Superiority; p = 0.8952, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -13.1, 90% CI 2-sided [-29.8 to 3.7], Standard Error of Mean 10.18
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 (Average Pain); Test type: Superiority; p = 0.1157, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 13.1, 90% CI 2-sided [-4.6 to 30.8], Standard Error of Mean 10.76
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 (Average Pain); Test type: Superiority; p = 0.4672, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 0.9, 90% CI 2-sided [-17.1 to 18.9], Standard Error of Mean 10.93
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 (Average Pain); Test type: Superiority; p = 0.9287, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -16.9, 90% CI 2-sided [-35.5 to 1.6], Standard Error of Mean 11.29
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 (Average Pain); Test type: Superiority; p = 0.4984, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 0.0, 90% CI 2-sided [-17.8 to 17.9], Standard Error of Mean 10.85
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 (Average Pain); Test type: Superiority; p = 0.9001, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -14.7, 90% CI 2-sided [-33.2 to 3.9], Standard Error of Mean 11.27
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 (Average Pain); Test type: Superiority; p = 0.8319, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -10.3, 90% CI 2-sided [-27.6 to 7.0], Standard Error of Mean 10.53
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 (Average Pain); Test type: Superiority; p = 0.0340, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 19.7, 90% CI 2-sided [2.3 to 37.0], Standard Error of Mean 10.55
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 (Average Pain); Test type: Superiority; p = 0.7359, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -6.8, 90% CI 2-sided [-24.4 to 10.8], Standard Error of Mean 10.70
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 (Average Pain); Test type: Superiority; p = 0.9291, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -16.0, 90% CI 2-sided [-33.3 to 1.3], Standard Error of Mean 10.51
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 (Average Pain); Test type: Superiority; p = 0.5087, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -0.2, 90% CI 2-sided [-17.4 to 16.9], Standard Error of Mean 10.44
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 (Average Pain); Test type: Superiority; p = 0.8098, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -9.5, 90% CI 2-sided [-27.2 to 8.1], Standard Error of Mean 10.74
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 (Average Pain); Test type: Superiority; p = 0.8114, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = -8.8, 90% CI 2-sided [-24.8 to 7.2], Standard Error of Mean 9.76
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 (Average Pain); Test type: Superiority; p = 0.1531, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 10.8, 90% CI 2-sided [-6.4 to 28.0], Standard Error of Mean 10.44
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 (Average Pain); Test type: Superiority; p = 0.3784, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 3.3, 90% CI 2-sided [-14.1 to 20.7], Standard Error of Mean 10.58

10. Secondary Outcome: Least Squares Mean of Percent Change From Baseline in PGA Skin Pain Numeric Rating Scale, at Worst, at Weeks 1, 2, 4, 6, 8, 12 and 16 -ANCOVA (FAS With Baseline ≥3, MI)
Description: Patient Global Assessment Skin Pain Numeric Rating Scale was used to assess the worst skin pain and the average skin pain due to HS. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). These two concepts were measured within the same instrument, but were scored separately. There was no composite score for this endpoint. The higher the score, the worse the outcomes, ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). Subscales were not combined. The ANCOVA model was fitted. Confidence interval (CI) was calculated using Blyth-Still-Casella method.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention with baseline ≥3 scores were included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 40 | 35 | 42 | 40
Percent change
  Week 1-Pain at its Worst | -1.45 [-9.33 to 6.42] | -8.89 [-17.18 to -0.61] | -11.97 [-19.58 to -4.37] | -15.58 [-23.50 to -7.66]
  Week 2-Pain at its Worst | -7.49 [-17.39 to 2.42] | -13.15 [-23.61 to -2.69] | -19.40 [-29.09 to -9.72] | -19.19 [-29.20 to -9.19]
  Week 4-Pain at its Worst | -18.81 [-29.31 to -8.31] | -15.56 [-26.68 to -4.45] | -26.63 [-36.88 to -16.37] | -19.98 [-30.63 to -9.33]
  Week 6-Pain at its Worst | -21.80 [-33.14 to -10.47] | -13.86 [-25.74 to -1.98] | -32.89 [-43.90 to -21.88] | -21.76 [-33.08 to -10.43]
  Week 8-Pain at its Worst | -23.53 [-34.49 to -12.57] | -20.70 [-32.22 to -9.18] | -34.83 [-45.55 to -24.11] | -23.37 [-34.40 to -12.35]
  Week 12-Pain at its Worst | -26.04 [-37.10 to -14.98] | -25.38 [-36.95 to -13.81] | -41.35 [-52.12 to -30.58] | -32.43 [-43.66 to -21.20]
  Week 16-Pain at its Worst | -22.34 [-33.82 to -10.86] | -19.77 [-31.60 to -7.93] | -43.88 [-55.06 to -32.70] | -34.87 [-46.36 to -23.38]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.1321, ANCOVA — One-sided p-value; Risk Difference (RD) = -7.44, 90% CI 2-sided [-18.39 to 3.52], Standard Error of Mean 6.661
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.0477, ANCOVA — One-sided p-value; Risk Difference (RD) = -10.52, 90% CI 2-sided [-20.90 to -0.14], Standard Error of Mean 6.308
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.0134, ANCOVA — One-sided p-value; Risk Difference (RD) = -14.13, 90% CI 2-sided [-24.62 to -3.63], Standard Error of Mean 6.379
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.2496, ANCOVA — One-sided p-value; Risk Difference (RD) = -5.66, 90% CI 2-sided [-19.45 to 8.12], Standard Error of Mean 8.380
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.0675, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.92, 90% CI 2-sided [-25.03 to 1.20], Standard Error of Mean 7.972
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.0730, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.71, 90% CI 2-sided [-24.96 to 1.54], Standard Error of Mean 8.054
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.6426, ANCOVA — One-sided p-value; Risk Difference (RD) = 3.25, 90% CI 2-sided [-11.38 to 17.88], Standard Error of Mean 8.892
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.1776, ANCOVA — One-sided p-value; Risk Difference (RD) = -7.82, 90% CI 2-sided [-21.73 to 6.09], Standard Error of Mean 8.457
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.4458, ANCOVA — One-sided p-value; Risk Difference (RD) = -1.17, 90% CI 2-sided [-15.28 to 12.94], Standard Error of Mean 8.579
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.7969, ANCOVA — One-sided p-value; Risk Difference (RD) = 7.94, 90% CI 2-sided [-7.79 to 23.68], Standard Error of Mean 9.566
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.1120, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.09, 90% CI 2-sided [-26.09 to 3.91], Standard Error of Mean 9.120
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.5021, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.05, 90% CI 2-sided [-15.06 to 15.16], Standard Error of Mean 9.188
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.6197, ANCOVA — One-sided p-value; Risk Difference (RD) = 2.83, 90% CI 2-sided [-12.46 to 18.12], Standard Error of Mean 9.296
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.1003, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.30, 90% CI 2-sided [-25.81 to 3.22], Standard Error of Mean 8.825
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.5070, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.16, 90% CI 2-sided [-14.50 to 14.81], Standard Error of Mean 8.908
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.5283, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.67, 90% CI 2-sided [-14.74 to 16.08], Standard Error of Mean 9.368
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.0431, ANCOVA — One-sided p-value; Risk Difference (RD) = -15.31, 90% CI 2-sided [-29.98 to -0.63], Standard Error of Mean 8.921
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.2395, ANCOVA — One-sided p-value; Risk Difference (RD) = -6.39, 90% CI 2-sided [-21.22 to 8.45], Standard Error of Mean 9.020
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.6054, ANCOVA — One-sided p-value; Risk Difference (RD) = 2.57, 90% CI 2-sided [-13.25 to 18.39], Standard Error of Mean 9.617
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.0106, ANCOVA — One-sided p-value; Risk Difference (RD) = -21.54, 90% CI 2-sided [-36.91 to -6.17], Standard Error of Mean 9.344
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.0890, ANCOVA — One-sided p-value; Risk Difference (RD) = -12.54, 90% CI 2-sided [-27.84 to 2.77], Standard Error of Mean 9.305

11. Secondary Outcome: Least Squares Mean of Percent Change From Baseline in PGA Skin Pain Numeric Rating Scale, on Average, at Weeks 1, 2, 4, 6, 8, 12 and 16 -ANCOVA (FAS With Baseline ≥3, MI)
Description: as for outcome 10
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention with baseline ≥3 scores were included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 38 | 32 | 41 | 34
Percent change
  Week 1-Average Pain | -2.47 [-9.45 to 4.51] | -8.64 [-16.06 to -1.22] | -13.53 [-20.29 to -6.77] | -8.81 [-16.53 to -1.10]
  Week 2-Average Pain | -11.24 [-19.66 to -2.83] | -13.39 [-22.42 to -4.37] | -21.59 [-29.80 to -13.38] | -13.49 [-22.78 to -4.20]
  Week 4-Average Pain | -24.04 [-34.14 to -13.94] | -16.00 [-26.79 to -5.21] | -33.01 [-42.90 to -23.13] | -18.67 [-29.57 to -7.77]
  Week 6-Average Pain | -28.65 [-39.19 to -18.10] | -14.86 [-26.11 to -3.61] | -38.04 [-48.30 to -27.77] | -22.60 [-34.04 to -11.16]
  Week 8-Average Pain | -30.75 [-41.20 to -20.31] | -21.78 [-32.86 to -10.70] | -39.59 [-49.80 to -29.39] | -22.11 [-33.48 to -10.75]
  Week 12-Average Pain | -30.85 [-40.83 to -20.87] | -28.50 [-39.14 to -17.87] | -45.24 [-54.97 to -35.50] | -30.42 [-41.28 to -19.57]
  Week 16-Average Pain | -27.83 [-37.98 to -17.69] | -23.80 [-34.41 to -13.18] | -46.21 [-56.05 to -36.37] | -31.92 [-42.93 to -20.91]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.1505, ANCOVA — One-sided p-value; Risk Difference (RD) = -6.17, 90% CI 2-sided [-15.98 to 3.64], Standard Error of Mean 5.963
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.0233, ANCOVA — One-sided p-value; Risk Difference (RD) = -11.06, 90% CI 2-sided [-20.19 to -1.92], Standard Error of Mean 5.555
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.1423, ANCOVA — One-sided p-value; Risk Difference (RD) = -6.34, 90% CI 2-sided [-16.09 to 3.41], Standard Error of Mean 5.926
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.3827, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.15, 90% CI 2-sided [-14.00 to 9.70], Standard Error of Mean 7.202
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.0624, ANCOVA — One-sided p-value; Risk Difference (RD) = -10.35, 90% CI 2-sided [-21.44 to 0.74], Standard Error of Mean 6.741
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.3771, ANCOVA — One-sided p-value; Risk Difference (RD) = -2.25, 90% CI 2-sided [-14.04 to 9.55], Standard Error of Mean 7.171
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.8247, ANCOVA — One-sided p-value; Risk Difference (RD) = 8.04, 90% CI 2-sided [-6.13 to 22.21], Standard Error of Mean 8.614
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.1337, ANCOVA — One-sided p-value; Risk Difference (RD) = -8.97, 90% CI 2-sided [-22.28 to 4.33], Standard Error of Mean 8.090
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.7357, ANCOVA — One-sided p-value; Risk Difference (RD) = 5.37, 90% CI 2-sided [-8.65 to 19.39], Standard Error of Mean 8.523
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.9377, ANCOVA — One-sided p-value; Risk Difference (RD) = 13.78, 90% CI 2-sided [-0.98 to 28.55], Standard Error of Mean 8.977
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.1332, ANCOVA — One-sided p-value; Risk Difference (RD) = -9.39, 90% CI 2-sided [-23.29 to 4.51], Standard Error of Mean 8.450
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.7514, ANCOVA — One-sided p-value; Risk Difference (RD) = 6.05, 90% CI 2-sided [-8.60 to 20.70], Standard Error of Mean 8.907
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.8433, ANCOVA — One-sided p-value; Risk Difference (RD) = 8.97, 90% CI 2-sided [-5.67 to 23.62], Standard Error of Mean 8.902
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.1461, ANCOVA — One-sided p-value; Risk Difference (RD) = -8.84, 90% CI 2-sided [-22.64 to 4.96], Standard Error of Mean 8.392
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.8364, ANCOVA — One-sided p-value; Risk Difference (RD) = 8.64, 90% CI 2-sided [-5.86 to 23.15], Standard Error of Mean 8.818
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.6085, ANCOVA — One-sided p-value; Risk Difference (RD) = 2.35, 90% CI 2-sided [-11.68 to 16.37], Standard Error of Mean 8.527
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.0365, ANCOVA — One-sided p-value; Risk Difference (RD) = -14.38, 90% CI 2-sided [-27.58 to -1.19], Standard Error of Mean 8.022
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.5201, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.43, 90% CI 2-sided [-13.50 to 14.36], Standard Error of Mean 8.469
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.6813, ANCOVA — One-sided p-value; Risk Difference (RD) = 4.04, 90% CI 2-sided [-10.05 to 18.12], Standard Error of Mean 8.564
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.0128, ANCOVA — One-sided p-value; Risk Difference (RD) = -18.38, 90% CI 2-sided [-31.91 to -4.84], Standard Error of Mean 8.230
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.3181, ANCOVA — One-sided p-value; Risk Difference (RD) = -4.09, 90% CI 2-sided [-18.30 to 10.12], Standard Error of Mean 8.639

12. Secondary Outcome: Least Squares Mean of Change From Baseline in PGA Skin Pain Numeric Rating Scale, at Worst, at Weeks 1, 2, 4, 6, 8, 12 and 16 - ANCOVA (FAS, MI)
Description: as for outcome 10
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 46 | 44 | 50 | 44
Percent change
  Week 1-Pain at its Worst | -0.23 [-0.59 to 0.13] | -0.54 [-0.91 to -0.16] | -0.68 [-1.03 to -0.33] | -0.71 [-1.09 to -0.33]
  Week 2-Pain at its Worst | -0.52 [-0.98 to -0.05] | -0.84 [-1.32 to -0.36] | -1.07 [-1.52 to -0.62] | -0.91 [-1.40 to -0.43]
  Week 4-Pain at its Worst | -1.22 [-1.74 to -0.70] | -1.15 [-1.68 to -0.61] | -1.67 [-2.17 to -1.16] | -1.19 [-1.74 to -0.65]
  Week 6-Pain at its Worst | -1.55 [-2.10 to -1.01] | -1.06 [-1.62 to -0.50] | -1.97 [-2.50 to -1.45] | -1.43 [-2.00 to -0.87]
  Week 8-Pain at its Worst | -1.56 [-2.11 to -1.01] | -1.40 [-1.97 to -0.83] | -1.95 [-2.48 to -1.41] | -1.43 [-2.01 to -0.86]
  Week 12-Pain at its Worst | -1.80 [-2.35 to -1.26] | -1.74 [-2.30 to -1.18] | -2.37 [-2.89 to -1.84] | -1.80 [-2.37 to -1.23]
  Week 16-Pain at its Worst | -1.44 [-2.00 to -0.89] | -1.35 [-1.91 to -0.80] | -2.51 [-3.04 to -1.98] | -2.01 [-2.58 to -1.44]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.1536, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.31, 90% CI 2-sided [-0.80 to 0.19], Standard Error of Mean 0.301
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.0581, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.45, 90% CI 2-sided [-0.93 to 0.02], Standard Error of Mean 0.289
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 Pain at its Worst; Test type: Superiority; p = 0.0532, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.48, 90% CI 2-sided [-0.98 to 0.01], Standard Error of Mean 0.300
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.2007, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.32, 90% CI 2-sided [-0.95 to 0.31], Standard Error of Mean 0.383
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.0694, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.55, 90% CI 2-sided [-1.16 to 0.06], Standard Error of Mean 0.370
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 Pain at its Worst; Test type: Superiority; p = 0.1509, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.39, 90% CI 2-sided [-1.02 to 0.23], Standard Error of Mean 0.382
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.5663, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.07, 90% CI 2-sided [-0.64 to 0.78], Standard Error of Mean 0.431
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.1396, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.45, 90% CI 2-sided [-1.13 to 0.23], Standard Error of Mean 0.416
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 Pain at its Worst; Test type: Superiority; p = 0.5227, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.02, 90% CI 2-sided [-0.69 to 0.74], Standard Error of Mean 0.432
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.8656, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.50, 90% CI 2-sided [-0.24 to 1.24], Standard Error of Mean 0.450
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.1671, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.42, 90% CI 2-sided [-1.13 to 0.29], Standard Error of Mean 0.434
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 Pain at its Worst; Test type: Superiority; p = 0.6063, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.62 to 0.86], Standard Error of Mean 0.450
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.6402, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.59 to 0.92], Standard Error of Mean 0.458
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.1916, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.38, 90% CI 2-sided [-1.11 to 0.34], Standard Error of Mean 0.441
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 Pain at its Worst; Test type: Superiority; p = 0.6119, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.13, 90% CI 2-sided [-0.62 to 0.88], Standard Error of Mean 0.456
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.5568, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.06, 90% CI 2-sided [-0.68 to 0.80], Standard Error of Mean 0.450
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.0976, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.56, 90% CI 2-sided [-1.27 to 0.15], Standard Error of Mean 0.433
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 Pain at its Worst; Test type: Superiority; p = 0.5001, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.00, 90% CI 2-sided [-0.74 to 0.74], Standard Error of Mean 0.451
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.5810, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.65 to 0.83], Standard Error of Mean 0.451
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.0079, ANCOVA — One-sided p-value; Risk Difference (RD) = -1.07, 90% CI 2-sided [-1.80 to -0.34], Standard Error of Mean 0.442
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 Pain at its Worst; Test type: Superiority; p = 0.1068, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.57, 90% CI 2-sided [-1.31 to 0.18], Standard Error of Mean 0.455

13. Secondary Outcome: Least Squares Mean of Change From Baseline in PGA Skin Pain Numeric Rating Scale, on Average, at Weeks 1, 2, 4, 6, 8, 12 and 16 - ANCOVA (FAS, MI)
Description: as for outcome 10
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 46 | 44 | 50 | 44
Percent change
  Week 1-Average Pain | -0.19 [-0.53 to 0.15] | -0.44 [-0.79 to -0.09] | -0.62 [-0.96 to -0.29] | -0.50 [-0.86 to -0.14]
  Week 2-Average Pain | -0.49 [-0.90 to -0.07] | -0.77 [-1.20 to -0.34] | -0.94 [-1.35 to -0.54] | -0.66 [-1.09 to -0.22]
  Week 4-Average Pain | -1.22 [-1.72 to -0.73] | -1.10 [-1.61 to -0.60] | -1.73 [-2.21 to -1.25] | -1.02 [-1.53 to -0.51]
  Week 6-Average Pain | -1.49 [-2.01 to -0.98] | -0.98 [-1.52 to -0.45] | -1.92 [-2.42 to -1.42] | -1.29 [-1.83 to -0.75]
  Week 8-Average Pain | -1.56 [-2.09 to -1.02] | -1.35 [-1.89 to -0.80] | -1.88 [-2.39 to -1.37] | -1.30 [-1.85 to -0.74]
  Week 12-Average Pain | -1.68 [-2.20 to -1.17] | -1.71 [-2.23 to -1.18] | -2.25 [-2.75 to -1.76] | -1.53 [-2.06 to -1.00]
  Week 16-Average Pain | -1.40 [-1.93 to -0.87] | -1.37 [-1.89 to -0.84] | -2.29 [-2.79 to -1.79] | -1.77 [-2.31 to -1.23]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.1898, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.25, 90% CI 2-sided [-0.72 to 0.22], Standard Error of Mean 0.284
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.0562, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.43, 90% CI 2-sided [-0.88 to 0.02], Standard Error of Mean 0.273
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1 Average Pain; Test type: Superiority; p = 0.1382, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.31, 90% CI 2-sided [-0.78 to 0.16], Standard Error of Mean 0.284
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.2039, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.28, 90% CI 2-sided [-0.85 to 0.28], Standard Error of Mean 0.343
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.0855, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.45, 90% CI 2-sided [-1.00 to 0.09], Standard Error of Mean 0.332
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2 Average Pain; Test type: Superiority; p = 0.3089, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.74 to 0.39], Standard Error of Mean 0.344
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.6124, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.55 to 0.79], Standard Error of Mean 0.407
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.1003, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.50, 90% CI 2-sided [-1.15 to 0.14], Standard Error of Mean 0.395
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4 Average Pain; Test type: Superiority; p = 0.6875, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.20, 90% CI 2-sided [-0.47 to 0.87], Standard Error of Mean 0.408
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.8833, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.51, 90% CI 2-sided [-0.19 to 1.21], Standard Error of Mean 0.427
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.1502, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.43, 90% CI 2-sided [-1.11 to 0.25], Standard Error of Mean 0.413
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6 Average Pain; Test type: Superiority; p = 0.6788, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.20, 90% CI 2-sided [-0.50 to 0.90], Standard Error of Mean 0.428
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.6835, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.21, 90% CI 2-sided [-0.51 to 0.94], Standard Error of Mean 0.441
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.2237, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.32, 90% CI 2-sided [-1.02 to 0.38], Standard Error of Mean 0.425
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8 Average Pain; Test type: Superiority; p = 0.7234, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.26, 90% CI 2-sided [-0.46 to 0.98], Standard Error of Mean 0.439
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.4773, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.72 to 0.67], Standard Error of Mean 0.424
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.0818, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.57, 90% CI 2-sided [-1.25 to 0.10], Standard Error of Mean 0.410
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12 Average Pain; Test type: Superiority; p = 0.6397, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.15, 90% CI 2-sided [-0.55 to 0.85], Standard Error of Mean 0.424
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.5321, ANCOVA — One-sided p-value; Risk Difference (RD) = 0.03, 90% CI 2-sided [-0.67 to 0.74], Standard Error of Mean 0.428
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.0167, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.89, 90% CI 2-sided [-1.59 to -0.20], Standard Error of Mean 0.420
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16 Average Pain; Test type: Superiority; p = 0.1963, ANCOVA — One-sided p-value; Risk Difference (RD) = -0.37, 90% CI 2-sided [-1.09 to 0.34], Standard Error of Mean 0.434

14. Secondary Outcome: Percentage of Participants Achieving Erythema Response Among Participants With Baseline Erythema Score ≥2 in at Least 1 Region at Weeks 1, 2, 4, 6, 8, 12 and 16 - MR (FAS, NRI)
Description: Erythema response was defined as achieving erythema score of 1 or 0 in all affected anatomic regions among participants who had an erythema score of 2 or more in at least 1 anatomic region at baseline. NRI for missing values which were related to withdrawal and all other events except for COVID-19. A four-point ordinal scale ranging was used: 0 (no redness), 1 (faint but discernible pink coloration), 2 (moderate red coloration), and 3 (very red or bright red coloration).
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention with baseline erythema score ≥2 scores in at least 1 region were included.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percentage of participants
  Week 1: number analyzed (Participants) | 46 | 43 | 46 | 44
  Week 1 | 6.5 [2.4 to 15.8] | 4.7 [1.2 to 13.2] | 8.7 [3.8 to 17.6] | 13.6 [6.1 to 24.3]
  Week 2: number analyzed (Participants) | 46 | 43 | 45 | 44
  Week 2 | 10.9 [5.4 to 21.3] | 20.9 [12.3 to 33.3] | 17.8 [9.2 to 29.7] | 18.2 [9.4 to 30.0]
  Week 4: number analyzed (Participants) | 45 | 43 | 46 | 44
  Week 4 | 13.3 [6.0 to 23.7] | 20.9 [12.3 to 33.3] | 28.3 [17.6 to 40.4] | 18.2 [9.4 to 30.0]
  Week 6: number analyzed (Participants) | 46 | 43 | 46 | 43
  Week 6 | 13.0 [5.8 to 23.2] | 27.9 [17.0 to 39.9] | 23.9 [15.1 to 35.0] | 23.3 [13.2 to 35.5]
  Week 8: number analyzed (Participants) | 46 | 43 | 46 | 43
  Week 8 | 15.2 [8.2 to 25.5] | 25.6 [16.3 to 37.7] | 28.3 [17.6 to 40.4] | 23.3 [13.2 to 35.5]
  Week 12: number analyzed (Participants) | 46 | 43 | 46 | 43
  Week 12 | 15.2 [8.2 to 25.5] | 23.3 [13.2 to 35.5] | 30.4 [20.4 to 43.4] | 18.6 [9.6 to 30.2]
  Week 16: number analyzed (Participants) | 46 | 43 | 46 | 43
  Week 16 | 13.0 [5.8 to 23.2] | 16.3 [8.8 to 27.0] | 28.3 [17.6 to 40.4] | 18.6 [9.6 to 30.2]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = -2.2, 90% CI 2-sided [-10.3 to 6.0], Standard Error of Mean 4.98
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = 2.0, 90% CI 2-sided [-7.3 to 11.3], Standard Error of Mean 5.64
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1; Test type: Superiority; Risk Difference (RD) = 6.8, 90% CI 2-sided [-3.9 to 17.4], Standard Error of Mean 6.47
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 10.7, 90% CI 2-sided [-2.0 to 23.4], Standard Error of Mean 7.74
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 7.6, 90% CI 2-sided [-4.5 to 19.7], Standard Error of Mean 7.34
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2; Test type: Superiority; Risk Difference (RD) = 7.5, 90% CI 2-sided [-4.6 to 19.6], Standard Error of Mean 7.36
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 7.4, 90% CI 2-sided [-5.7 to 20.5], Standard Error of Mean 7.95
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 15.1, 90% CI 2-sided [1.4 to 28.7], Standard Error of Mean 8.33
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 4.8, 90% CI 2-sided [-8.0 to 17.5], Standard Error of Mean 7.74
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 14.3, 90% CI 2-sided [0.7 to 28.0], Standard Error of Mean 8.30
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 10.9, 90% CI 2-sided [-2.2 to 24.0], Standard Error of Mean 7.96
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6; Test type: Superiority; Risk Difference (RD) = 10.6, 90% CI 2-sided [-2.6 to 23.9], Standard Error of Mean 8.06
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; p = 0.1162, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 10.1, 90% CI 2-sided [-3.6 to 23.9], Standard Error of Mean 8.38
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; p = 0.0642, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 13.1, 90% CI 2-sided [-0.8 to 27.0], Standard Error of Mean 8.43
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; p = 0.1664, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 8.1, 90% CI 2-sided [-5.7 to 21.8], Standard Error of Mean 8.36
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; p = 0.1882, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 7.2, 90% CI 2-sided [-6.1 to 20.5], Standard Error of Mean 8.10
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; p = 0.0423, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 14.9, 90% CI 2-sided [1.1 to 28.8], Standard Error of Mean 8.43
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; p = 0.3396, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 3.3, 90% CI 2-sided [-9.7 to 16.3], Standard Error of Mean 7.90
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; p = 0.3584, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 2.7, 90% CI 2-sided [-9.4 to 14.8], Standard Error of Mean 7.35
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; p = 0.0367, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 14.9, 90% CI 2-sided [1.5 to 28.3], Standard Error of Mean 8.17
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; p = 0.2486, MR weighting strategy — One-sided p-value; P-value method for risk difference (RD) was minimum risk (MR) weighting strategy by Mehrotra and Railkar (2000); Risk Difference (RD) = 5.2, 90% CI 2-sided [-7.4 to 17.8], Standard Error of Mean 7.65

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: The treatment-emergent AEs (TEAEs) were considered as an adverse event that started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time was flagged as TEAEs.
Time Frame: Up to 20 weeks
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Participants
  Participants with adverse events | 23 | 26 | 30 | 29
  Participants with serious adverse events | 0 | 2 | 0 | 2
  Participants with severe adverse events | 1 | 2 | 1 | 4
  Participants discontinued from study due to adverse events | 0 | 1 | 1 | 6
  Participants discontinued study drug due to AE and continued Study | 1 | 2 | 2 | 1
  Participants with temporary discontinuation due to adverse events | 2 | 1 | 3 | 5

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related)
Description: as for outcome 15
Time Frame: Up to 20 weeks
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Participants
  Participants with adverse events | 7 | 10 | 12 | 16
  Participants with serious adverse events | 0 | 1 | 0 | 1
  Participants with severe adverse events | 0 | 1 | 0 | 3
  Participants discontinued from study due to adverse events | 0 | 1 | 1 | 4
  Participants discontinued study drug due to AE and continued Study | 1 | 1 | 2 | 0
  Participants with temporary discontinuation due to adverse events | 1 | 1 | 0 | 2

17. Secondary Outcome: Number of Participants With Incidence of Post-baseline Vital Signs of Clinical Concern - Increase From Baseline (Safety Analysis Set)
Description: The vital signs were measured included temperature (Oral, Tympanic, Axillary or Temporal), pulse rate (beats/min) and blood pressure (mmHg).
Time Frame: Up to 20 weeks
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Participants
  Supine Diastolic Blood Pressure (MMHG): Change >= 20mmHg increase | 2 | 1 | 2 | 4
  Supine Systolic Blood Pressure (MMHG): Change >= 30mmHg increase | 1 | 1 | 2 | 4

18. Secondary Outcome: Number of Participants With Incidence of Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) (Safety Analysis Set)
Description: Laboratory test abnormalities included hematology, chemistry, urinalysis and biomarker.
Time Frame: Up to 20 weeks
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Participants
  Hematology: hemoglobin (g/dL) <0.8x lower limit of normal (LLN): number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: hemoglobin (g/dL) <0.8x lower limit of normal (LLN) | 1 | 0 | 4 | 0
  Hematology: Hematocrit (%) <0.8x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Hematocrit (%) <0.8x LLN | 0 | 0 | 1 | 0
  Hematology: Erythrocytes (10^6/mm^3) <0.8x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Erythrocytes (10^6/mm^3) <0.8x LLN | 0 | 0 | 3 | 1
  Hematology: Ery. Mean Corpuscular Volume (um^3) <0.9x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular Volume (um^3) <0.9x LLN | 1 | 2 | 1 | 0
  Hematology: Ery. Mean Corpuscular Volume (um^3) >1.1x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular Volume (um^3) >1.1x ULN | 0 | 2 | 1 | 1
  Hematology: Ery. Mean Corpuscular Hemoglobin (pg/cell) <0.9x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular Hemoglobin (pg/cell) <0.9x LLN | 5 | 5 | 7 | 5
  Hematology: Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1x ULN | 0 | 0 | 0 | 0
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9x LLN | 6 | 3 | 6 | 6
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1x ULN | 0 | 0 | 0 | 0
  Hematology: Mean Platelet Volume (fL) <0.9x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Mean Platelet Volume (fL) <0.9x LLN | 0 | 0 | 0 | 2
  Hematology: Mean Platelet Volume (fL) >1.1x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Mean Platelet Volume (fL) >1.1x ULN | 1 | 0 | 0 | 0
  Hematology: Platelets (10^3/mm^3) <0.5x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Platelets (10^3/mm^3) <0.5x LLN | 0 | 0 | 0 | 1
  Hematology: Platelets (10^3/mm^3) >1.75x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Platelets (10^3/mm^3) >1.75x ULN | 0 | 0 | 1 | 3
  Hematology: Leukocytes (10^3/mm^3) <0.6x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Leukocytes (10^3/mm^3) <0.6x LLN | 0 | 0 | 1 | 3
  Hematology: Leukocytes (10^3/mm^3) >1.5x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Leukocytes (10^3/mm^3) >1.5x ULN | 4 | 1 | 1 | 0
  Hematology: Lymphocytes (10^3/mm^3) <0.8x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Lymphocytes (10^3/mm^3) <0.8x LLN | 1 | 0 | 1 | 3
  Hematology: Lymphocytes (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Lymphocytes (10^3/mm^3) >1.2x ULN | 5 | 2 | 7 | 4
  Hematology: Neutrophils (10^3/mm^3) <0.8x LLN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Neutrophils (10^3/mm^3) <0.8x LLN | 0 | 0 | 3 | 8
  Hematology: Neutrophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Neutrophils (10^3/mm^3) >1.2x ULN | 8 | 3 | 6 | 4
  Hematology: Basophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Basophils (10^3/mm^3) >1.2x ULN | 0 | 0 | 0 | 0
  Hematology: Eosinophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Eosinophils (10^3/mm^3) >1.2x ULN | 0 | 1 | 0 | 0
  Hematology: Monocytes (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 47 | 46 | 52 | 47
  Hematology: Monocytes (10^3/mm^3) >1.2x ULN | 2 | 0 | 0 | 0
  Clinical Chemistry: Bilirubin (mg/dL) >1.5x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Aspartate Aminotransferase (U/L) >3.0x ULN | 0 | 1 | 1 | 0
  Clinical Chemistry: Alanine Aminotransferase (U/L) >3.0x ULN | 0 | 1 | 2 | 1
  Clinical Chemistry: Alkaline Phosphatase (U/L) >3.0x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Protein (g/dL) <0.8x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Protein (g/dL) >1.2x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Albumin (g/dL) <0.8x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Albumin (g/dL) >1.2x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Urea Nitrogen (mg/dL) >1.3x ULN | 0 | 1 | 0 | 2
  Clinical Chemistry: Creatinine (mg/dL) >1.3x ULN | 0 | 0 | 1 | 0
  Clinical Chemistry: Urate (mg/dL) >1.2x ULN | 3 | 3 | 4 | 6
  Clinical Chemistry: Cholesterol (mg/dL) >1.3x ULN: number analyzed (Participants) | 41 | 39 | 45 | 37
  Clinical Chemistry: Cholesterol (mg/dL) >1.3x ULN | 2 | 1 | 4 | 2
  Clinical Chemistry: HDL Cholesterol (mg/dL) <0.8x LLN: number analyzed (Participants) | 41 | 39 | 45 | 37
  Clinical Chemistry: HDL Cholesterol (mg/dL) <0.8x LLN | 10 | 6 | 6 | 5
  Clinical Chemistry: LDL Cholesterol (mg/dL) >1.2x ULN: number analyzed (Participants) | 41 | 39 | 45 | 37
  Clinical Chemistry: LDL Cholesterol (mg/dL) >1.2x ULN | 1 | 1 | 3 | 2
  Clinical Chemistry: Triglycerides (mg/dL) >1.3x ULN: number analyzed (Participants) | 41 | 39 | 45 | 37
  Clinical Chemistry: Triglycerides (mg/dL) >1.3x ULN | 5 | 4 | 6 | 7
  Clinical Chemistry: Sodium (mEq/L) <0.95x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Sodium (mEq/L) >1.05x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Potassium (mEq/L) <0.9x LLN | 1 | 1 | 1 | 0
  Clinical Chemistry: Potassium (mEq/L) >1.1x ULN | 1 | 2 | 0 | 2
  Clinical Chemistry: Chloride (mEq/L) <0.9x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Chloride (mEq/L) >1.1x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Calcium (mg/dL) <0.9x LLN | 0 | 2 | 0 | 0
  Clinical Chemistry: Calcium (mg/dL) >1.1x ULN | 0 | 0 | 0 | 0
  Clinical Chemistry: Bicarbonate (mEq/L) <0.9x LLN | 10 | 10 | 2 | 13
  Clinical Chemistry: Bicarbonate (mEq/L) >1.1x ULN | 0 | 1 | 0 | 0
  Clinical Chemistry: Glucose (mg/dL) <0.6x LLN: number analyzed (Participants) | 31 | 28 | 31 | 33
  Clinical Chemistry: Glucose (mg/dL) <0.6x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Glucose (mg/dL) >1.5x ULN: number analyzed (Participants) | 31 | 28 | 31 | 33
  Clinical Chemistry: Glucose (mg/dL) >1.5x ULN | 1 | 2 | 1 | 3
  Clinical Chemistry: Creatine Kinase (U/L) >2.0x ULN | 6 | 2 | 18 | 20
  Clinical Chemistry: Glucose -FASTING (mg/dL) <0.6x LLN: number analyzed (Participants) | 46 | 44 | 49 | 43
  Clinical Chemistry: Glucose -FASTING (mg/dL) <0.6x LLN | 0 | 0 | 0 | 0
  Clinical Chemistry: Glucose -FASTING (mg/dL) >1.5x ULN: number analyzed (Participants) | 46 | 44 | 49 | 43
  Clinical Chemistry: Glucose -FASTING (mg/dL) >1.5x ULN | 4 | 5 | 3 | 5
  Urinalysis: pH <4.5 | 0 | 0 | 0 | 0
  Urinalysis: pH >8 | 2 | 1 | 2 | 5
  Urinalysis: URINE Glucose (mg/dL) ≥1 | 4 | 6 | 2 | 4
  Urinalysis: Ketones (mg/dL) ≥1 | 9 | 6 | 8 | 12
  Urinalysis: URINE Protein (mg/dL) ≥1 | 32 | 30 | 29 | 32
  Urinalysis: URINE Hemoglobin ≥1 | 23 | 9 | 16 | 10
  Urinalysis: Urobilinogen (EU/dL) ≥1 | 3 | 4 | 7 | 5
  Urinalysis: URINE Bilirubin ≥1 | 0 | 0 | 0 | 0
  Urinalysis: Nitrite ≥1 | 3 | 4 | 6 | 3
  Urinalysis: Leukocyte Esterase ≥1 | 10 | 5 | 9 | 6
  Urinalysis: URINE Erythrocytes (/HPF) ≥20: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: URINE Erythrocytes (/HPF) ≥20 | 4 | 2 | 5 | 1
  Urinalysis: Granular Casts (/LPF) >1: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: Granular Casts (/LPF) >1 | 0 | 0 | 0 | 0
  Urinalysis: Hyaline Casts (/LPF) >1: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: Hyaline Casts (/LPF) >1 | 1 | 1 | 1 | 2
  Urinalysis: RBC Casts (/LPF) >1: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: RBC Casts (/LPF) >1 | 0 | 0 | 0 | 0
  Urinalysis: WBC Casts (/LPF) >1: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: WBC Casts (/LPF) >1 | 0 | 0 | 0 | 0
  Urinalysis: Bacteria (/HPF) >20: number analyzed (Participants) | 44 | 36 | 42 | 39
  Urinalysis: Bacteria (/HPF) >20 | 6 | 6 | 5 | 4
  Biomarker: C Reactive Protein (mg/dL) >1.1x ULN: number analyzed (Participants) | 47 | 46 | 52 | 45
  Biomarker: C Reactive Protein (mg/dL) >1.1x ULN | 37 | 29 | 37 | 30

19. Secondary Outcome: Number of Participants With Incidence of Post-baseline Electrocardiogram (ECG) Values of Clinical Concern (Safety Analysis Set)
Description: ECG parameters included QT interval, QTc interval, PR interval, and QRS complex.
Time Frame: Up to 20 weeks
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention with post-baseline result. If participants didn't have any post-baseline measurement, the participants were not included in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 47 | 45 | 50 | 45
Participants
  PR INTERVAL, SINGLE BEAT (MSEC): Value>280 | 0 | 0 | 0 | 0
  QRS DURATION, SINGLE BEAT (MSEC): Value>120 | 2 | 0 | 3 | 1
  QT INTERVAL, SINGLE BEAT (MSEC): Value>500 | 0 | 0 | 0 | 0
  QTCB INTERVAL, SINGLE BEAT (MSEC): 450<Value<=480 | 12 | 12 | 16 | 7
  QTCB INTERVAL, SINGLE BEAT (MSEC): 480<Value<500 | 1 | 0 | 2 | 1
  QTCB INTERVAL, SINGLE BEAT (MSEC): Value>=500 | 1 | 0 | 1 | 0
  QTCB INTERVAL, SINGLE BEAT (MSEC): 30<=Chg<=60 | 9 | 12 | 13 | 6
  QTCB INTERVAL, SINGLE BEAT (MSEC): Chg>60 | 0 | 1 | 1 | 0
  QTCF INTERVAL, SINGLE BEAT (MSEC): 450<Value<=480 | 2 | 2 | 6 | 2
  QTCF INTERVAL, SINGLE BEAT (MSEC): 480<Value<500 | 1 | 0 | 1 | 0
  QTCF INTERVAL, SINGLE BEAT (MSEC): Value>=500 | 0 | 0 | 0 | 0
  QTCF INTERVAL, SINGLE BEAT (MSEC): 30<=Chg<=60 | 5 | 6 | 7 | 2
  QTCF INTERVAL, SINGLE BEAT (MSEC): Chg>60 | 0 | 1 | 1 | 0

20. Secondary Outcome: Least Squares Mean of Absolute Score in Hidradenitis Suppurativa (HS) Symptom Items up to Week 16 - Mixed Effect Model Repeated Measurement (MMRM) (FAS, OBS)
Description: The Hidradenitis Suppurativa Symptom Items were 5 single items that assessed patient self-reported symptoms related to HS. The participants were asked to rate each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom. The symptoms assessed include: pain, tenderness, swelling, tiredness, and bother of lesion appearance. The higher the score, the worse the outcomes, ranging from 0 indicating no symptom experience and 10 indicating the worst possible symptom. These concepts were scored separately, and were not combined into a composite score. When using mixed effect model repeated measurement (MMRM) analysis, only observed data were used and missing data were not imputed.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Units on a scale
  Week 1-HSS0101-Pain At It's Worst: number analyzed (Participants) | 48 | 46 | 51 | 45
  Week 1-HSS0101-Pain At It's Worst | 5.67 [5.33 to 6.01] | 5.47 [5.13 to 5.82] | 5.19 [4.86 to 5.52] | 5.25 [4.90 to 5.60]
  Week 2-HSS0101-Pain At It's Worst: number analyzed (Participants) | 48 | 42 | 50 | 43
  Week 2-HSS0101-Pain At It's Worst | 5.39 [4.95 to 5.84] | 5.10 [4.63 to 5.57] | 4.69 [4.25 to 5.12] | 4.83 [4.36 to 5.29]
  Week 4-HSS0101-Pain At It's Worst: number analyzed (Participants) | 46 | 37 | 47 | 39
  Week 4-HSS0101-Pain At It's Worst | 4.75 [4.21 to 5.29] | 5.01 [4.42 to 5.59] | 4.36 [3.83 to 4.89] | 4.69 [4.11 to 5.26]
  Week 6-HSS0101-Pain At It's Worst: number analyzed (Participants) | 45 | 38 | 44 | 36
  Week 6-HSS0101-Pain At It's Worst | 4.39 [3.80 to 4.98] | 5.02 [4.38 to 5.65] | 4.20 [3.61 to 4.79] | 4.60 [3.96 to 5.24]
  Week 8-HSS0101-Pain At It's Worst: number analyzed (Participants) | 42 | 37 | 44 | 32
  Week 8-HSS0101-Pain At It's Worst | 4.46 [3.83 to 5.09] | 4.70 [4.02 to 5.37] | 4.14 [3.51 to 4.77] | 4.91 [4.22 to 5.60]
  Week 12-HSS0101-Pain At It's Worst: number analyzed (Participants) | 36 | 28 | 35 | 29
  Week 12-HSS0101-Pain At It's Worst | 4.28 [3.63 to 4.92] | 4.44 [3.73 to 5.15] | 3.60 [2.95 to 4.24] | 4.35 [3.65 to 5.06]
  Week 16-HSS0101-Pain At It's Worst: number analyzed (Participants) | 28 | 25 | 32 | 25
  Week 16-HSS0101-Pain At It's Worst | 4.77 [4.06 to 5.48] | 4.86 [4.09 to 5.62] | 3.53 [2.83 to 4.22] | 3.87 [3.11 to 4.62]
  Week 1-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 48 | 46 | 51 | 45
  Week 1-HSS0102-Tenderness At It's Worst | 5.66 [5.33 to 5.99] | 5.66 [5.32 to 6.00] | 5.37 [5.05 to 5.69] | 5.35 [5.01 to 5.69]
  Week 2-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 48 | 42 | 50 | 43
  Week 2-HSS0102-Tenderness At It's Worst | 5.46 [5.05 to 5.87] | 5.24 [4.81 to 5.67] | 5.06 [4.66 to 5.46] | 5.00 [4.57 to 5.43]
  Week 4-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 46 | 37 | 47 | 39
  Week 4-HSS0102-Tenderness At It's Worst | 4.85 [4.33 to 5.38] | 5.07 [4.50 to 5.65] | 4.61 [4.09 to 5.13] | 4.75 [4.18 to 5.31]
  Week 6-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 45 | 38 | 44 | 36
  Week 6-HSS0102-Tenderness At It's Worst | 4.65 [4.06 to 5.23] | 5.12 [4.49 to 5.75] | 4.41 [3.82 to 5.00] | 4.65 [4.02 to 5.29]
  Week 8-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 42 | 37 | 44 | 32
  Week 8-HSS0102-Tenderness At It's Worst | 4.69 [4.08 to 5.31] | 4.78 [4.13 to 5.44] | 4.45 [3.84 to 5.06] | 5.04 [4.37 to 5.71]
  Week 12-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 36 | 28 | 35 | 29
  Week 12-HSS0102-Tenderness At It's Worst | 4.40 [3.78 to 5.01] | 4.45 [3.77 to 5.13] | 3.90 [3.29 to 4.52] | 4.41 [3.74 to 5.09]
  Week 16-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 28 | 25 | 32 | 25
  Week 16-HSS0102-Tenderness At It's Worst | 5.04 [4.36 to 5.73] | 5.08 [4.35 to 5.82] | 3.80 [3.14 to 4.47] | 3.93 [3.20 to 4.66]
  Week 1-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 48 | 46 | 51 | 45
  Week 1-HSS0103-Swelling At It's Worst | 5.53 [5.20 to 5.86] | 5.43 [5.09 to 5.77] | 5.30 [4.98 to 5.62] | 5.07 [4.73 to 5.40]
  Week 2-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 48 | 42 | 50 | 43
  Week 2-HSS0103-Swelling At It's Worst | 5.17 [4.76 to 5.58] | 4.93 [4.50 to 5.36] | 4.70 [4.31 to 5.10] | 4.77 [4.35 to 5.20]
  Week 4-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 46 | 37 | 47 | 39
  Week 4-HSS0103-Swelling At It's Worst | 4.57 [4.07 to 5.07] | 4.73 [4.19 to 5.27] | 4.40 [3.91 to 4.89] | 4.66 [4.12 to 5.19]
  Week 6-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 45 | 38 | 44 | 36
  Week 6-HSS0103-Swelling At It's Worst | 4.36 [3.79 to 4.94] | 5.06 [4.44 to 5.68] | 4.35 [3.77 to 4.92] | 4.60 [3.97 to 5.22]
  Week 8-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 42 | 37 | 44 | 32
  Week 8-HSS0103-Swelling At It's Worst | 4.38 [3.81 to 4.96] | 4.67 [4.06 to 5.28] | 4.38 [3.81 to 4.96] | 4.88 [4.26 to 5.51]
  Week 12-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 36 | 28 | 35 | 29
  Week 12-HSS0103-Swelling At It's Worst | 4.34 [3.75 to 4.93] | 4.40 [3.75 to 5.06] | 3.87 [3.28 to 4.47] | 4.30 [3.65 to 4.95]
  Week 16-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 28 | 25 | 32 | 25
  Week 16-HSS0103-Swelling At It's Worst | 4.79 [4.12 to 5.45] | 5.02 [4.30 to 5.73] | 3.73 [3.08 to 4.37] | 3.77 [3.06 to 4.47]
  Week 1-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 48 | 46 | 51 | 45
  Week 1-HSS0104-Tiredness At It's Worst | 5.55 [5.24 to 5.85] | 5.71 [5.40 to 6.02] | 4.98 [4.68 to 5.27] | 5.63 [5.32 to 5.94]
  Week 2-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 48 | 42 | 50 | 43
  Week 2-HSS0104-Tiredness At It's Worst | 5.10 [4.69 to 5.51] | 5.16 [4.73 to 5.58] | 4.66 [4.26 to 5.06] | 5.36 [4.94 to 5.79]
  Week 4-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 46 | 37 | 47 | 39
  Week 4-HSS0104-Tiredness At It's Worst | 5.05 [4.56 to 5.54] | 4.93 [4.41 to 5.46] | 4.24 [3.76 to 4.72] | 4.91 [4.39 to 5.42]
  Week 6-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 45 | 38 | 44 | 36
  Week 6-HSS0104-Tiredness At It's Worst | 4.77 [4.23 to 5.32] | 4.81 [4.23 to 5.40] | 4.25 [3.71 to 4.80] | 4.89 [4.30 to 5.48]
  Week 8-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 42 | 37 | 44 | 32
  Week 8-HSS0104-Tiredness At It's Worst | 4.86 [4.31 to 5.41] | 4.69 [4.11 to 5.28] | 4.32 [3.78 to 4.87] | 4.97 [4.38 to 5.56]
  Week 12-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 36 | 28 | 35 | 29
  Week 12-HSS0104-Tiredness At It's Worst | 4.80 [4.21 to 5.38] | 4.46 [3.81 to 5.10] | 3.99 [3.40 to 4.57] | 4.95 [4.30 to 5.59]
  Week 16-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 28 | 25 | 32 | 25
  Week 16-HSS0104-Tiredness At It's Worst | 4.59 [3.96 to 5.22] | 4.81 [4.14 to 5.49] | 4.03 [3.42 to 4.65] | 4.68 [4.01 to 5.36]
  Week 1-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 48 | 46 | 51 | 45
  Week 1-HSS0105-Bothered By Appearance HS Lesion | 7.38 [7.08 to 7.69] | 7.43 [7.12 to 7.75] | 7.06 [6.76 to 7.36] | 7.37 [7.05 to 7.68]
  Week 2-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 48 | 42 | 50 | 43
  Week 2-HSS0105-Bothered By Appearance HS Lesion | 7.34 [6.96 to 7.72] | 7.24 [6.84 to 7.64] | 6.55 [6.18 to 6.92] | 6.99 [6.59 to 7.38]
  Week 4-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 46 | 37 | 47 | 39
  Week 4-HSS0105-Bothered By Appearance HS Lesion | 6.94 [6.48 to 7.41] | 7.26 [6.77 to 7.76] | 6.00 [5.54 to 6.46] | 6.65 [6.16 to 7.15]
  Week 6-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 45 | 38 | 44 | 36
  Week 6-HSS0105-Bothered By Appearance HS Lesion | 6.69 [6.18 to 7.21] | 7.24 [6.69 to 7.79] | 6.00 [5.49 to 6.52] | 6.59 [6.04 to 7.15]
  Week 8-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 42 | 37 | 44 | 32
  Week 8-HSS0105-Bothered By Appearance HS Lesion | 6.98 [6.42 to 7.53] | 6.82 [6.23 to 7.41] | 5.86 [5.31 to 6.42] | 6.67 [6.07 to 7.28]
  Week 12-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 36 | 28 | 35 | 29
  Week 12-HSS0105-Bothered By Appearance HS Lesion | 6.46 [5.84 to 7.07] | 6.51 [5.84 to 7.17] | 5.59 [4.98 to 6.20] | 6.58 [5.91 to 7.24]
  Week 16-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 28 | 25 | 32 | 25
  Week 16-HSS0105-Bothered By Appearance HS Lesion | 6.37 [5.69 to 7.05] | 6.77 [6.04 to 7.50] | 5.43 [4.76 to 6.09] | 6.37 [5.64 to 7.09]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.20, 90% CI 2-sided [-0.69 to 0.29], Standard Error of Mean 0.295
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.48, 90% CI 2-sided [-0.96 to -0.01], Standard Error of Mean 0.287
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.42, 90% CI 2-sided [-0.91 to 0.06], Standard Error of Mean 0.295
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.30, 90% CI 2-sided [-0.95 to 0.35], Standard Error of Mean 0.392
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.71, 90% CI 2-sided [-1.33 to -0.08], Standard Error of Mean 0.377
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.57, 90% CI 2-sided [-1.21 to 0.08], Standard Error of Mean 0.391
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.26, 90% CI 2-sided [-0.54 to 1.05], Standard Error of Mean 0.481
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.39, 90% CI 2-sided [-1.15 to 0.37], Standard Error of Mean 0.458
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.06, 90% CI 2-sided [-0.85 to 0.73], Standard Error of Mean 0.478
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.62, 90% CI 2-sided [-0.24 to 1.49], Standard Error of Mean 0.524
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.19, 90% CI 2-sided [-1.03 to 0.64], Standard Error of Mean 0.505
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.21, 90% CI 2-sided [-0.66 to 1.08], Standard Error of Mean 0.526
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.24, 90% CI 2-sided [-0.69 to 1.16], Standard Error of Mean 0.558
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.32, 90% CI 2-sided [-1.21 to 0.57], Standard Error of Mean 0.539
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.44, 90% CI 2-sided [-0.49 to 1.38], Standard Error of Mean 0.565
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.79 to 1.12], Standard Error of Mean 0.578
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.68, 90% CI 2-sided [-1.59 to 0.23], Standard Error of Mean 0.550
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.88 to 1.03], Standard Error of Mean 0.576
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.96 to 1.13], Standard Error of Mean 0.631
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.25, 90% CI 2-sided [-2.24 to -0.25], Standard Error of Mean 0.600
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.91, 90% CI 2-sided [-1.95 to 0.13], Standard Error of Mean 0.628
Statistical Analysis 22: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.01, 90% CI 2-sided [-0.47 to 0.48], Standard Error of Mean 0.286
Statistical Analysis 23: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.28, 90% CI 2-sided [-0.75 to 0.18], Standard Error of Mean 0.278
Statistical Analysis 24: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.31, 90% CI 2-sided [-0.78 to 0.17], Standard Error of Mean 0.286
Statistical Analysis 25: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.22, 90% CI 2-sided [-0.81 to 0.38], Standard Error of Mean 0.361
Statistical Analysis 26: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.40, 90% CI 2-sided [-0.97 to 0.18], Standard Error of Mean 0.347
Statistical Analysis 27: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.46, 90% CI 2-sided [-1.05 to 0.14], Standard Error of Mean 0.360
Statistical Analysis 28: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [-0.56 to 1.00], Standard Error of Mean 0.471
Statistical Analysis 29: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.25, 90% CI 2-sided [-0.99 to 0.49], Standard Error of Mean 0.448
Statistical Analysis 30: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.11, 90% CI 2-sided [-0.88 to 0.67], Standard Error of Mean 0.468
Statistical Analysis 31: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.48, 90% CI 2-sided [-0.38 to 1.34], Standard Error of Mean 0.520
Statistical Analysis 32: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.23, 90% CI 2-sided [-1.06 to 0.60], Standard Error of Mean 0.501
Statistical Analysis 33: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.01, 90% CI 2-sided [-0.86 to 0.87], Standard Error of Mean 0.523
Statistical Analysis 34: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.81 to 0.99], Standard Error of Mean 0.542
Statistical Analysis 35: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.25, 90% CI 2-sided [-1.11 to 0.62], Standard Error of Mean 0.523
Statistical Analysis 36: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.35, 90% CI 2-sided [-0.56 to 1.25], Standard Error of Mean 0.549
Statistical Analysis 37: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.87 to 0.97], Standard Error of Mean 0.554
Statistical Analysis 38: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.49, 90% CI 2-sided [-1.36 to 0.38], Standard Error of Mean 0.527
Statistical Analysis 39: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.02, 90% CI 2-sided [-0.90 to 0.93], Standard Error of Mean 0.552
Statistical Analysis 40: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.96 to 1.04], Standard Error of Mean 0.606
Statistical Analysis 41: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.24, 90% CI 2-sided [-2.19 to -0.29], Standard Error of Mean 0.577
Statistical Analysis 42: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.11, 90% CI 2-sided [-2.11 to -0.11], Standard Error of Mean 0.603
Statistical Analysis 43: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.57 to 0.37], Standard Error of Mean 0.284
Statistical Analysis 44: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.23, 90% CI 2-sided [-0.69 to 0.22], Standard Error of Mean 0.278
Statistical Analysis 45: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.47, 90% CI 2-sided [-0.94 to 0.01], Standard Error of Mean 0.285
Statistical Analysis 46: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.24, 90% CI 2-sided [-0.83 to 0.35], Standard Error of Mean 0.357
Statistical Analysis 47: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.46, 90% CI 2-sided [-1.03 to 0.11], Standard Error of Mean 0.345
Statistical Analysis 48: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.40, 90% CI 2-sided [-0.99 to 0.19], Standard Error of Mean 0.357
Statistical Analysis 49: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.58 to 0.90], Standard Error of Mean 0.446
Statistical Analysis 50: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.87 to 0.53], Standard Error of Mean 0.424
Statistical Analysis 51: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.65 to 0.82], Standard Error of Mean 0.443
Statistical Analysis 52: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.70, 90% CI 2-sided [-0.15 to 1.54], Standard Error of Mean 0.510
Statistical Analysis 53: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.83 to 0.80], Standard Error of Mean 0.493
Statistical Analysis 54: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [-0.62 to 1.08], Standard Error of Mean 0.513
Statistical Analysis 55: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.29, 90% CI 2-sided [-0.55 to 1.13], Standard Error of Mean 0.507
Statistical Analysis 56: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.00, 90% CI 2-sided [-0.81 to 0.81], Standard Error of Mean 0.489
Statistical Analysis 57: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.50, 90% CI 2-sided [-0.35 to 1.35], Standard Error of Mean 0.514
Statistical Analysis 58: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.07, 90% CI 2-sided [-0.81 to 0.95], Standard Error of Mean 0.532
Statistical Analysis 59: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.47, 90% CI 2-sided [-1.30 to 0.37], Standard Error of Mean 0.505
Statistical Analysis 60: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.04, 90% CI 2-sided [-0.92 to 0.84], Standard Error of Mean 0.530
Statistical Analysis 61: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [-0.75 to 1.20], Standard Error of Mean 0.589
Statistical Analysis 62: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.06, 90% CI 2-sided [-1.99 to -0.13], Standard Error of Mean 0.561
Statistical Analysis 63: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.02, 90% CI 2-sided [-1.99 to -0.05], Standard Error of Mean 0.586
Statistical Analysis 64: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.27 to 0.59], Standard Error of Mean 0.262
Statistical Analysis 65: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.57, 90% CI 2-sided [-0.99 to -0.15], Standard Error of Mean 0.255
Statistical Analysis 66: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.35 to 0.52], Standard Error of Mean 0.262
Statistical Analysis 67: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.06, 90% CI 2-sided [-0.54 to 0.65], Standard Error of Mean 0.357
Statistical Analysis 68: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.44, 90% CI 2-sided [-1.01 to 0.13], Standard Error of Mean 0.344
Statistical Analysis 69: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.26, 90% CI 2-sided [-0.33 to 0.85], Standard Error of Mean 0.356
Statistical Analysis 70: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.12, 90% CI 2-sided [-0.83 to 0.60], Standard Error of Mean 0.434
Statistical Analysis 71: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.81, 90% CI 2-sided [-1.49 to -0.12], Standard Error of Mean 0.414
Statistical Analysis 72: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.14, 90% CI 2-sided [-0.86 to 0.57], Standard Error of Mean 0.431
Statistical Analysis 73: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.76 to 0.84], Standard Error of Mean 0.483
Statistical Analysis 74: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.52, 90% CI 2-sided [-1.29 to 0.26], Standard Error of Mean 0.466
Statistical Analysis 75: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.68 to 0.92], Standard Error of Mean 0.485
Statistical Analysis 76: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.96 to 0.63], Standard Error of Mean 0.483
Statistical Analysis 77: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.53, 90% CI 2-sided [-1.31 to 0.24], Standard Error of Mean 0.466
Statistical Analysis 78: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.11, 90% CI 2-sided [-0.69 to 0.92], Standard Error of Mean 0.488
Statistical Analysis 79: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.34, 90% CI 2-sided [-1.21 to 0.53], Standard Error of Mean 0.527
Statistical Analysis 80: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.81, 90% CI 2-sided [-1.64 to 0.02], Standard Error of Mean 0.503
Statistical Analysis 81: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.15, 90% CI 2-sided [-0.72 to 1.02], Standard Error of Mean 0.527
Statistical Analysis 82: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [-0.70 to 1.15], Standard Error of Mean 0.559
Statistical Analysis 83: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.56, 90% CI 2-sided [-1.44 to 0.32], Standard Error of Mean 0.532
Statistical Analysis 84: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.83 to 1.01], Standard Error of Mean 0.557
Statistical Analysis 85: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.39 to 0.49], Standard Error of Mean 0.264
Statistical Analysis 86: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.32, 90% CI 2-sided [-0.75 to 0.10], Standard Error of Mean 0.257
Statistical Analysis 87: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.46 to 0.42], Standard Error of Mean 0.266
Statistical Analysis 88: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.65 to 0.45], Standard Error of Mean 0.333
Statistical Analysis 89: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.80, 90% CI 2-sided [-1.33 to -0.27], Standard Error of Mean 0.321
Statistical Analysis 90: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.36, 90% CI 2-sided [-0.91 to 0.19], Standard Error of Mean 0.333
Statistical Analysis 91: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.32, 90% CI 2-sided [-0.36 to 1.00], Standard Error of Mean 0.411
Statistical Analysis 92: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.94, 90% CI 2-sided [-1.59 to -0.29], Standard Error of Mean 0.393
Statistical Analysis 93: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.29, 90% CI 2-sided [-0.97 to 0.39], Standard Error of Mean 0.411
Statistical Analysis 94: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.55, 90% CI 2-sided [-0.20 to 1.30], Standard Error of Mean 0.454
Statistical Analysis 95: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.69, 90% CI 2-sided [-1.41 to 0.04], Standard Error of Mean 0.439
Statistical Analysis 96: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.85 to 0.66], Standard Error of Mean 0.456
Statistical Analysis 97: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.15, 90% CI 2-sided [-0.96 to 0.66], Standard Error of Mean 0.491
Statistical Analysis 98: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -1.11, 90% CI 2-sided [-1.89 to -0.33], Standard Error of Mean 0.473
Statistical Analysis 99: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.30, 90% CI 2-sided [-1.13 to 0.52], Standard Error of Mean 0.497
Statistical Analysis 100: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.86 to 0.95], Standard Error of Mean 0.547
Statistical Analysis 101: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.87, 90% CI 2-sided [-1.73 to -0.01], Standard Error of Mean 0.523
Statistical Analysis 102: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.78 to 1.03], Standard Error of Mean 0.547
Statistical Analysis 103: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.39, 90% CI 2-sided [-0.60 to 1.39], Standard Error of Mean 0.602
Statistical Analysis 104: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.95, 90% CI 2-sided [-1.90 to 0.00], Standard Error of Mean 0.574
Statistical Analysis 105: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.01, 90% CI 2-sided [-1.00 to 0.99], Standard Error of Mean 0.600

21. Secondary Outcome: Least Squares Mean of Change From Baseline in Hidradenitis Suppurativa (HS) Symptom Items up to Week 16 - MMRM (FAS, OBS)
Description: as for outcome 20
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Units on a scale
  Week 1-HSS0101-Pain At It's Worst: number analyzed (Participants) | 47 | 45 | 50 | 45
  Week 1-HSS0101-Pain At It's Worst | -0.19 [-0.53 to 0.15] | -0.39 [-0.74 to -0.04] | -0.67 [-1.00 to -0.34] | -0.61 [-0.96 to -0.26]
  Week 2-HSS0101-Pain At It's Worst: number analyzed (Participants) | 47 | 41 | 49 | 42
  Week 2-HSS0101-Pain At It's Worst | -0.47 [-0.92 to -0.02] | -0.77 [-1.24 to -0.30] | -1.18 [-1.61 to -0.74] | -1.04 [-1.50 to -0.57]
  Week 4-HSS0101-Pain At It's Worst: number analyzed (Participants) | 46 | 36 | 47 | 38
  Week 4-HSS0101-Pain At It's Worst | -1.12 [-1.66 to -0.58] | -0.86 [-1.44 to -0.27] | -1.51 [-2.04 to -0.98] | -1.18 [-1.76 to -0.60]
  Week 6-HSS0101-Pain At It's Worst: number analyzed (Participants) | 45 | 37 | 42 | 36
  Week 6-HSS0101-Pain At It's Worst | -1.47 [-2.06 to -0.88] | -0.85 [-1.48 to -0.21] | -1.66 [-2.26 to -1.07] | -1.27 [-1.91 to -0.63]
  Week 8-HSS0101-Pain At It's Worst: number analyzed (Participants) | 42 | 36 | 42 | 32
  Week 8-HSS0101-Pain At It's Worst | -1.40 [-2.03 to -0.77] | -1.17 [-1.84 to -0.49] | -1.72 [-2.35 to -1.09] | -0.96 [-1.65 to -0.27]
  Week 12-HSS0101-Pain At It's Worst: number analyzed (Participants) | 36 | 27 | 34 | 28
  Week 12-HSS0101-Pain At It's Worst | -1.59 [-2.23 to -0.94] | -1.42 [-2.13 to -0.72] | -2.27 [-2.91 to -1.62] | -1.51 [-2.21 to -0.81]
  Week 16-HSS0101-Pain At It's Worst: number analyzed (Participants) | 28 | 24 | 30 | 25
  Week 16-HSS0101-Pain At It's Worst | -1.09 [-1.80 to -0.38] | -1.01 [-1.77 to -0.24] | -2.34 [-3.03 to -1.64] | -2.00 [-2.75 to -1.24]
  Week 1-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 47 | 45 | 50 | 45
  Week 1-HSS0102-Tenderness At It's Worst | -0.37 [-0.70 to -0.04] | -0.36 [-0.70 to -0.02] | -0.65 [-0.97 to -0.33] | -0.67 [-1.01 to -0.33]
  Week 2-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 47 | 41 | 49 | 42
  Week 2-HSS0102-Tenderness At It's Worst | -0.56 [-0.97 to -0.15] | -0.78 [-1.21 to -0.35] | -0.96 [-1.36 to -0.56] | -1.02 [-1.45 to -0.59]
  Week 4-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 46 | 36 | 47 | 38
  Week 4-HSS0102-Tenderness At It's Worst | -1.17 [-1.70 to -0.64] | -0.95 [-1.52 to -0.37] | -1.42 [-1.94 to -0.90] | -1.28 [-1.84 to -0.71]
  Week 6-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 45 | 37 | 42 | 36
  Week 6-HSS0102-Tenderness At It's Worst | -1.38 [-1.96 to -0.79] | -0.90 [-1.53 to -0.27] | -1.61 [-2.20 to -1.02] | -1.37 [-2.00 to -0.73]
  Week 8-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 42 | 36 | 42 | 32
  Week 8-HSS0102-Tenderness At It's Worst | -1.33 [-1.94 to -0.72] | -1.24 [-1.89 to -0.58] | -1.58 [-2.19 to -0.96] | -0.98 [-1.65 to -0.31]
  Week 12-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 36 | 27 | 34 | 28
  Week 12-HSS0102-Tenderness At It's Worst | -1.63 [-2.24 to -1.01] | -1.57 [-2.25 to -0.90] | -2.12 [-2.74 to -1.50] | -1.61 [-2.28 to -0.93]
  Week 16-HSS0102-Tenderness At It's Worst: number analyzed (Participants) | 28 | 24 | 30 | 25
  Week 16-HSS0102-Tenderness At It's Worst | -0.98 [-1.66 to -0.30] | -0.94 [-1.67 to -0.20] | -2.22 [-2.89 to -1.55] | -2.09 [-2.82 to -1.36]
  Week 1-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 47 | 45 | 50 | 45
  Week 1-HSS0103-Swelling At It's Worst | -0.24 [-0.56 to 0.09] | -0.34 [-0.67 to 0.00] | -0.47 [-0.79 to -0.15] | -0.70 [-1.04 to -0.36]
  Week 2-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 47 | 41 | 49 | 42
  Week 2-HSS0103-Swelling At It's Worst | -0.60 [-1.01 to -0.19] | -0.84 [-1.27 to -0.41] | -1.06 [-1.46 to -0.66] | -1.00 [-1.42 to -0.57]
  Week 4-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 46 | 36 | 47 | 38
  Week 4-HSS0103-Swelling At It's Worst | -1.20 [-1.70 to -0.70] | -1.04 [-1.58 to -0.50] | -1.37 [-1.86 to -0.87] | -1.11 [-1.65 to -0.57]
  Week 6-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 45 | 37 | 42 | 36
  Week 6-HSS0103-Swelling At It's Worst | -1.40 [-1.98 to -0.83] | -0.71 [-1.33 to -0.09] | -1.42 [-2.00 to -0.84] | -1.17 [-1.80 to -0.55]
  Week 8-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 42 | 36 | 42 | 32
  Week 8-HSS0103-Swelling At It's Worst | -1.38 [-1.96 to -0.81] | -1.10 [-1.71 to -0.48] | -1.38 [-1.96 to -0.81] | -0.88 [-1.51 to -0.26]
  Week 12-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 36 | 27 | 34 | 28
  Week 12-HSS0103-Swelling At It's Worst | -1.43 [-2.02 to -0.84] | -1.36 [-2.02 to -0.71] | -1.90 [-2.49 to -1.30] | -1.47 [-2.12 to -0.82]
  Week 16-HSS0103-Swelling At It's Worst: number analyzed (Participants) | 28 | 24 | 30 | 25
  Week 16-HSS0103-Swelling At It's Worst | -0.98 [-1.64 to -0.32] | -0.75 [-1.47 to -0.04] | -2.04 [-2.69 to -1.39] | -2.00 [-2.71 to -1.29]
  Week 1-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 47 | 45 | 50 | 45
  Week 1-HSS0104-Tiredness At It's Worst | -0.04 [-0.34 to 0.26] | 0.12 [-0.19 to 0.43] | -0.61 [-0.91 to -0.32] | 0.04 [-0.26 to 0.35]
  Week 2-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 47 | 41 | 49 | 42
  Week 2-HSS0104-Tiredness At It's Worst | -0.49 [-0.90 to -0.08] | -0.43 [-0.86 to -0.01] | -0.93 [-1.32 to -0.53] | -0.23 [-0.65 to 0.20]
  Week 4-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 46 | 36 | 47 | 38
  Week 4-HSS0104-Tiredness At It's Worst | -0.54 [-1.03 to -0.05] | -0.66 [-1.18 to -0.13] | -1.35 [-1.83 to -0.87] | -0.68 [-1.20 to -0.16]
  Week 6-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 45 | 37 | 42 | 36
  Week 6-HSS0104-Tiredness At It's Worst | -0.82 [-1.36 to -0.27] | -0.78 [-1.36 to -0.19] | -1.33 [-1.88 to -0.79] | -0.70 [-1.29 to -0.11]
  Week 8-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 42 | 36 | 42 | 32
  Week 8-HSS0104-Tiredness At It's Worst | -0.73 [-1.28 to -0.18] | -0.90 [-1.48 to -0.31] | -1.26 [-1.81 to -0.72] | -0.62 [-1.21 to -0.02]
  Week 12-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 36 | 27 | 34 | 28
  Week 12-HSS0104-Tiredness At It's Worst | -0.79 [-1.38 to -0.20] | -1.13 [-1.77 to -0.49] | -1.60 [-2.19 to -1.02] | -0.64 [-1.28 to 0.00]
  Week 16-HSS0104-Tiredness At It's Worst: number analyzed (Participants) | 28 | 24 | 30 | 25
  Week 16-HSS0104-Tiredness At It's Worst | -1.00 [-1.63 to -0.37] | -0.78 [-1.45 to -0.10] | -1.56 [-2.17 to -0.94] | -0.90 [-1.58 to -0.23]
  Week 1-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 47 | 45 | 50 | 45
  Week 1-HSS0105-Bothered By Appearance HS Lesion | -0.19 [-0.49 to 0.12] | -0.14 [-0.45 to 0.18] | -0.51 [-0.81 to -0.21] | -0.20 [-0.52 to 0.11]
  Week 2-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 47 | 41 | 49 | 42
  Week 2-HSS0105-Bothered By Appearance HS Lesion | -0.23 [-0.61 to 0.15] | -0.33 [-0.73 to 0.07] | -1.02 [-1.39 to -0.65] | -0.58 [-0.98 to -0.19]
  Week 4-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 46 | 36 | 47 | 38
  Week 4-HSS0105-Bothered By Appearance HS Lesion | -0.63 [-1.09 to -0.16] | -0.30 [-0.80 to 0.19] | -1.57 [-2.02 to -1.11] | -0.92 [-1.41 to -0.42]
  Week 6-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 45 | 37 | 42 | 36
  Week 6-HSS0105-Bothered By Appearance HS Lesion | -0.88 [-1.39 to -0.36] | -0.33 [-0.88 to 0.22] | -1.56 [-2.08 to -1.05] | -0.97 [-1.53 to -0.42]
  Week 8-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 42 | 36 | 42 | 32
  Week 8-HSS0105-Bothered By Appearance HS Lesion | -0.59 [-1.15 to -0.04] | -0.75 [-1.34 to -0.15] | -1.71 [-2.26 to -1.15] | -0.90 [-1.50 to -0.29]
  Week 12-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 36 | 27 | 34 | 28
  Week 12-HSS0105-Bothered By Appearance HS Lesion | -1.11 [-1.73 to -0.50] | -1.06 [-1.73 to -0.40] | -1.98 [-2.59 to -1.37] | -0.99 [-1.66 to -0.33]
  Week 16-HSS0105-Bothered By Appearance HS Lesion: number analyzed (Participants) | 28 | 24 | 30 | 25
  Week 16-HSS0105-Bothered By Appearance HS Lesion | -1.20 [-1.87 to -0.52] | -0.80 [-1.53 to -0.07] | -2.14 [-2.81 to -1.48] | -1.20 [-1.92 to -0.48]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.20, 90% CI 2-sided [-0.69 to 0.29], Standard Error of Mean 0.295
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.48, 90% CI 2-sided [-0.96 to -0.01], Standard Error of Mean 0.287
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.42, 90% CI 2-sided [-0.91 to 0.06], Standard Error of Mean 0.295
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.30, 90% CI 2-sided [-0.95 to 0.35], Standard Error of Mean 0.392
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.71, 90% CI 2-sided [-1.33 to -0.08], Standard Error of Mean 0.377
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.57, 90% CI 2-sided [-1.21 to 0.08], Standard Error of Mean 0.391
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.26, 90% CI 2-sided [-0.54 to 1.05], Standard Error of Mean 0.481
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.39, 90% CI 2-sided [-1.15 to 0.37], Standard Error of Mean 0.458
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.06, 90% CI 2-sided [-0.85 to 0.73], Standard Error of Mean 0.478
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.62, 90% CI 2-sided [-0.24 to 1.49], Standard Error of Mean 0.524
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.19, 90% CI 2-sided [-1.03 to 0.64], Standard Error of Mean 0.505
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.21, 90% CI 2-sided [-0.66 to 1.08], Standard Error of Mean 0.526
Statistical Analysis 13: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.24, 90% CI 2-sided [-0.69 to 1.16], Standard Error of Mean 0.558
Statistical Analysis 14: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.32, 90% CI 2-sided [-1.21 to 0.57], Standard Error of Mean 0.539
Statistical Analysis 15: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.44, 90% CI 2-sided [-0.49 to 1.38], Standard Error of Mean 0.565
Statistical Analysis 16: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.79 to 1.12], Standard Error of Mean 0.578
Statistical Analysis 17: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.68, 90% CI 2-sided [-1.59 to 0.23], Standard Error of Mean 0.550
Statistical Analysis 18: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.88 to 1.03], Standard Error of Mean 0.576
Statistical Analysis 19: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.96 to 1.13], Standard Error of Mean 0.631
Statistical Analysis 20: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.25, 90% CI 2-sided [-2.24 to -0.25], Standard Error of Mean 0.600
Statistical Analysis 21: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0101-Pain At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.91, 90% CI 2-sided [-1.95 to 0.13], Standard Error of Mean 0.628
Statistical Analysis 22: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.01, 90% CI 2-sided [-0.47 to 0.48], Standard Error of Mean 0.286
Statistical Analysis 23: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.28, 90% CI 2-sided [-0.75 to 0.18], Standard Error of Mean 0.278
Statistical Analysis 24: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.31, 90% CI 2-sided [-0.78 to 0.17], Standard Error of Mean 0.286
Statistical Analysis 25: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.22, 90% CI 2-sided [-0.81 to 0.38], Standard Error of Mean 0.361
Statistical Analysis 26: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.40, 90% CI 2-sided [-0.97 to 0.18], Standard Error of Mean 0.347
Statistical Analysis 27: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.46, 90% CI 2-sided [-1.05 to 0.14], Standard Error of Mean 0.360
Statistical Analysis 28: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [-0.56 to 1.00], Standard Error of Mean 0.471
Statistical Analysis 29: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.25, 90% CI 2-sided [-0.99 to 0.49], Standard Error of Mean 0.448
Statistical Analysis 30: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.11, 90% CI 2-sided [-0.88 to 0.67], Standard Error of Mean 0.468
Statistical Analysis 31: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.48, 90% CI 2-sided [-0.38 to 1.34], Standard Error of Mean 0.520
Statistical Analysis 32: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.23, 90% CI 2-sided [-1.06 to 0.60], Standard Error of Mean 0.501
Statistical Analysis 33: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.01, 90% CI 2-sided [-0.86 to 0.87], Standard Error of Mean 0.523
Statistical Analysis 34: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.81 to 0.99], Standard Error of Mean 0.542
Statistical Analysis 35: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.25, 90% CI 2-sided [-1.11 to 0.62], Standard Error of Mean 0.523
Statistical Analysis 36: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.35, 90% CI 2-sided [-0.56 to 1.25], Standard Error of Mean 0.549
Statistical Analysis 37: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.87 to 0.97], Standard Error of Mean 0.554
Statistical Analysis 38: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.49, 90% CI 2-sided [-1.36 to 0.38], Standard Error of Mean 0.527
Statistical Analysis 39: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.02, 90% CI 2-sided [-0.90 to 0.93], Standard Error of Mean 0.552
Statistical Analysis 40: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.96 to 1.04], Standard Error of Mean 0.606
Statistical Analysis 41: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.24, 90% CI 2-sided [-2.19 to -0.29], Standard Error of Mean 0.577
Statistical Analysis 42: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0102-Tenderness At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.11, 90% CI 2-sided [-2.11 to -0.11], Standard Error of Mean 0.603
Statistical Analysis 43: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.57 to 0.37], Standard Error of Mean 0.284
Statistical Analysis 44: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.23, 90% CI 2-sided [-0.69 to 0.22], Standard Error of Mean 0.278
Statistical Analysis 45: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.47, 90% CI 2-sided [-0.94 to 0.01], Standard Error of Mean 0.285
Statistical Analysis 46: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.24, 90% CI 2-sided [-0.83 to 0.35], Standard Error of Mean 0.357
Statistical Analysis 47: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.46, 90% CI 2-sided [-1.03 to 0.11], Standard Error of Mean 0.345
Statistical Analysis 48: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.40, 90% CI 2-sided [-0.99 to 0.19], Standard Error of Mean 0.357
Statistical Analysis 49: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.58 to 0.90], Standard Error of Mean 0.446
Statistical Analysis 50: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.87 to 0.53], Standard Error of Mean 0.424
Statistical Analysis 51: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.65 to 0.82], Standard Error of Mean 0.443
Statistical Analysis 52: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.70, 90% CI 2-sided [-0.15 to 1.54], Standard Error of Mean 0.510
Statistical Analysis 53: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.83 to 0.80], Standard Error of Mean 0.493
Statistical Analysis 54: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [-0.62 to 1.08], Standard Error of Mean 0.513
Statistical Analysis 55: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.29, 90% CI 2-sided [-0.55 to 1.13], Standard Error of Mean 0.507
Statistical Analysis 56: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.00, 90% CI 2-sided [-0.81 to 0.81], Standard Error of Mean 0.489
Statistical Analysis 57: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.50, 90% CI 2-sided [-0.35 to 1.35], Standard Error of Mean 0.514
Statistical Analysis 58: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.07, 90% CI 2-sided [-0.81 to 0.95], Standard Error of Mean 0.532
Statistical Analysis 59: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.47, 90% CI 2-sided [-1.30 to 0.37], Standard Error of Mean 0.505
Statistical Analysis 60: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.04, 90% CI 2-sided [-0.92 to 0.84], Standard Error of Mean 0.530
Statistical Analysis 61: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [-0.75 to 1.20], Standard Error of Mean 0.589
Statistical Analysis 62: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.06, 90% CI 2-sided [-1.99 to -0.13], Standard Error of Mean 0.561
Statistical Analysis 63: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0103-Swelling At It's Worst; Test type: Superiority; Risk Difference (RD) = -1.02, 90% CI 2-sided [-1.99 to -0.05], Standard Error of Mean 0.586
Statistical Analysis 64: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.27 to 0.59], Standard Error of Mean 0.262
Statistical Analysis 65: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.57, 90% CI 2-sided [-0.99 to -0.15], Standard Error of Mean 0.255
Statistical Analysis 66: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.35 to 0.52], Standard Error of Mean 0.262
Statistical Analysis 67: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.06, 90% CI 2-sided [-0.54 to 0.65], Standard Error of Mean 0.357
Statistical Analysis 68: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.44, 90% CI 2-sided [-1.01 to 0.13], Standard Error of Mean 0.344
Statistical Analysis 69: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.26, 90% CI 2-sided [-0.33 to 0.85], Standard Error of Mean 0.356
Statistical Analysis 70: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.12, 90% CI 2-sided [-0.83 to 0.60], Standard Error of Mean 0.434
Statistical Analysis 71: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.81, 90% CI 2-sided [-1.49 to -0.12], Standard Error of Mean 0.414
Statistical Analysis 72: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.14, 90% CI 2-sided [-0.86 to 0.57], Standard Error of Mean 0.431
Statistical Analysis 73: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.76 to 0.84], Standard Error of Mean 0.483
Statistical Analysis 74: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.52, 90% CI 2-sided [-1.29 to 0.26], Standard Error of Mean 0.466
Statistical Analysis 75: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.68 to 0.92], Standard Error of Mean 0.485
Statistical Analysis 76: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.96 to 0.63], Standard Error of Mean 0.483
Statistical Analysis 77: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.53, 90% CI 2-sided [-1.31 to 0.24], Standard Error of Mean 0.466
Statistical Analysis 78: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.11, 90% CI 2-sided [-0.69 to 0.92], Standard Error of Mean 0.488
Statistical Analysis 79: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.34, 90% CI 2-sided [-1.21 to 0.53], Standard Error of Mean 0.527
Statistical Analysis 80: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.81, 90% CI 2-sided [-1.64 to 0.02], Standard Error of Mean 0.503
Statistical Analysis 81: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.15, 90% CI 2-sided [-0.72 to 1.02], Standard Error of Mean 0.527
Statistical Analysis 82: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [-0.70 to 1.15], Standard Error of Mean 0.559
Statistical Analysis 83: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = -0.56, 90% CI 2-sided [-1.44 to 0.32], Standard Error of Mean 0.532
Statistical Analysis 84: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0104-Tiredness At It's Worst; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.83 to 1.01], Standard Error of Mean 0.557
Statistical Analysis 85: Comparison: Placebo vs PF-06650833 400mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.39 to 0.49], Standard Error of Mean 0.264
Statistical Analysis 86: Comparison: Placebo vs PF-06700841 45mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.32, 90% CI 2-sided [-0.75 to 0.10], Standard Error of Mean 0.257
Statistical Analysis 87: Comparison: Placebo vs PF-06826647 400mg QD; Week 1-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.46 to 0.42], Standard Error of Mean 0.266
Statistical Analysis 88: Comparison: Placebo vs PF-06650833 400mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.65 to 0.45], Standard Error of Mean 0.333
Statistical Analysis 89: Comparison: Placebo vs PF-06700841 45mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.80, 90% CI 2-sided [-1.33 to -0.27], Standard Error of Mean 0.321
Statistical Analysis 90: Comparison: Placebo vs PF-06826647 400mg QD; Week 2-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.36, 90% CI 2-sided [-0.91 to 0.19], Standard Error of Mean 0.333
Statistical Analysis 91: Comparison: Placebo vs PF-06650833 400mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.32, 90% CI 2-sided [-0.36 to 1.00], Standard Error of Mean 0.411
Statistical Analysis 92: Comparison: Placebo vs PF-06700841 45mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.94, 90% CI 2-sided [-1.59 to -0.29], Standard Error of Mean 0.393
Statistical Analysis 93: Comparison: Placebo vs PF-06826647 400mg QD; Week 4-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.29, 90% CI 2-sided [-0.97 to 0.39], Standard Error of Mean 0.411
Statistical Analysis 94: Comparison: Placebo vs PF-06650833 400mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.55, 90% CI 2-sided [-0.20 to 1.30], Standard Error of Mean 0.454
Statistical Analysis 95: Comparison: Placebo vs PF-06700841 45mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.69, 90% CI 2-sided [-1.41 to 0.04], Standard Error of Mean 0.439
Statistical Analysis 96: Comparison: Placebo vs PF-06826647 400mg QD; Week 6-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.85 to 0.66], Standard Error of Mean 0.456
Statistical Analysis 97: Comparison: Placebo vs PF-06650833 400mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.15, 90% CI 2-sided [-0.96 to 0.66], Standard Error of Mean 0.491
Statistical Analysis 98: Comparison: Placebo vs PF-06700841 45mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -1.11, 90% CI 2-sided [-1.89 to -0.33], Standard Error of Mean 0.473
Statistical Analysis 99: Comparison: Placebo vs PF-06826647 400mg QD; Week 8-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.30, 90% CI 2-sided [-1.13 to 0.52], Standard Error of Mean 0.497
Statistical Analysis 100: Comparison: Placebo vs PF-06650833 400mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.86 to 0.95], Standard Error of Mean 0.547
Statistical Analysis 101: Comparison: Placebo vs PF-06700841 45mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.87, 90% CI 2-sided [-1.73 to -0.01], Standard Error of Mean 0.523
Statistical Analysis 102: Comparison: Placebo vs PF-06826647 400mg QD; Week 12-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.78 to 1.03], Standard Error of Mean 0.547
Statistical Analysis 103: Comparison: Placebo vs PF-06650833 400mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = 0.39, 90% CI 2-sided [-0.60 to 1.39], Standard Error of Mean 0.602
Statistical Analysis 104: Comparison: Placebo vs PF-06700841 45mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.95, 90% CI 2-sided [-1.90 to 0.00], Standard Error of Mean 0.574
Statistical Analysis 105: Comparison: Placebo vs PF-06826647 400mg QD; Week 16-HSS0105-Bothered By Appearance HS Lesion; Test type: Superiority; Risk Difference (RD) = -0.01, 90% CI 2-sided [-1.00 to 0.99], Standard Error of Mean 0.600

22. Secondary Outcome: Least Squares Mean of Absolute Score in Dermatology Life Quality Index (DLQI) Total Score up to Week 16 - MMRM (FAS, OBS)
Description: The Dermatology Life Quality Index (DLQI) is a general dermatology questionnaire that consists of 10 items that assess patient health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment) over the last week. Scoring for each item is on a qualitative 0 to 3 scale, with options of "Not at all", "A little", "A lot", "Very much". The scores are added up to a total composite score with the range from the minimum score of 0 to the maximum score of 30. The higher the score, the worse the outcomes.
Time Frame: At weeks 4, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Units on a scale
  Week 4-Absolute Score: number analyzed (Participants) | 44 | 40 | 39 | 33
  Week 4-Absolute Score | 10.2 [8.6 to 11.7] | 10.6 [9.0 to 12.2] | 9.6 [8.1 to 11.2] | 11.1 [9.4 to 12.8]
  Week 8-Absolute Score: number analyzed (Participants) | 44 | 39 | 42 | 36
  Week 8-Absolute Score | 10.8 [9.3 to 12.3] | 10.2 [8.7 to 11.8] | 9.6 [8.1 to 11.2] | 10.8 [9.2 to 12.4]
  Week 12-Absolute Score: number analyzed (Participants) | 40 | 32 | 37 | 34
  Week 12-Absolute Score | 10.7 [9.1 to 12.3] | 9.9 [8.1 to 11.7] | 8.7 [7.1 to 10.4] | 10.5 [8.7 to 12.2]
  Week 16-Absolute Score: number analyzed (Participants) | 37 | 29 | 35 | 29
  Week 16-Absolute Score | 9.5 [7.8 to 11.1] | 11.2 [9.4 to 13.1] | 8.2 [6.5 to 10.0] | 9.5 [7.7 to 11.4]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 0.4, 90% CI 2-sided [-1.7 to 2.6], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -0.5, 90% CI 2-sided [-2.7 to 1.7], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 0.9, 90% CI 2-sided [-1.4 to 3.2], Standard Error of Mean 1.38
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = -0.5, 90% CI 2-sided [-2.7 to 1.6], Standard Error of Mean 1.31
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = -1.1, 90% CI 2-sided [-3.3 to 1.0], Standard Error of Mean 1.29
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = 0.0, 90% CI 2-sided [-2.2 to 2.2], Standard Error of Mean 1.34
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -0.8, 90% CI 2-sided [-3.2 to 1.6], Standard Error of Mean 1.44
Statistical Analysis 8: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -2.0, 90% CI 2-sided [-4.3 to 0.3], Standard Error of Mean 1.39
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -0.2, 90% CI 2-sided [-2.6 to 2.2], Standard Error of Mean 1.45
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 1.7, 90% CI 2-sided [-0.7 to 4.2], Standard Error of Mean 1.50
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = -1.2, 90% CI 2-sided [-3.6 to 1.2], Standard Error of Mean 1.45
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 0.1, 90% CI 2-sided [-2.4 to 2.6], Standard Error of Mean 1.51

23. Secondary Outcome: Least Squares Mean of Change From Baseline in DLQI Total Score up to Week 16 - MMRM (FAS, OBS)
Description: The Dermatology Life Quality Index (DLQI) is a general dermatology questionnaire that consists of 10 items that assess patient health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment) over the last week. Scoring for each item is on a qualitative 0 to 3 scale, with options of "Not at all", "A little", "A lot", "Very much". The scores are added up to a total composite score with the range from the minimum score of 0 to the maximum score of 30. The higher the score, the worse the outcomes. The assessments examined a change from baseline in total score, where negative value means improvement in DLQI.
Time Frame: At weeks 4, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Units on a scale
  Week 4-Change from Baseline: number analyzed (Participants) | 41 | 39 | 37 | 31
  Week 4-Change from Baseline | -5.5 [-7.1 to -4.0] | -5.1 [-6.7 to -3.5] | -6.1 [-7.6 to -4.5] | -4.6 [-6.3 to -2.9]
  Week 8-Change from Baseline: number analyzed (Participants) | 41 | 37 | 40 | 34
  Week 8-Change from Baseline | -4.9 [-6.4 to -3.4] | -5.5 [-7.0 to -3.9] | -6.1 [-7.6 to -4.5] | -4.9 [-6.5 to -3.3]
  Week 12-Change from Baseline: number analyzed (Participants) | 38 | 31 | 36 | 31
  Week 12-Change from Baseline | -5.0 [-6.6 to -3.4] | -5.8 [-7.6 to -4.0] | -6.9 [-8.6 to -5.3] | -5.2 [-7.0 to -3.5]
  Week 16-Change from Baseline: number analyzed (Participants) | 35 | 28 | 32 | 27
  Week 16-Change from Baseline | -6.2 [-7.9 to -4.5] | -4.5 [-6.3 to -2.6] | -7.5 [-9.2 to -5.7] | -6.2 [-8.0 to -4.3]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 0.4, 90% CI 2-sided [-1.7 to 2.6], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -0.5, 90% CI 2-sided [-2.7 to 1.7], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 0.9, 90% CI 2-sided [-1.4 to 3.2], Standard Error of Mean 1.38
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = -0.5, 90% CI 2-sided [-2.7 to 1.6], Standard Error of Mean 1.31
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = -1.1, 90% CI 2-sided [-3.3 to 1.0], Standard Error of Mean 1.29
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = 0.0, 90% CI 2-sided [-2.2 to 2.2], Standard Error of Mean 1.34
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -0.8, 90% CI 2-sided [-3.2 to 1.6], Standard Error of Mean 1.44
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -2.0, 90% CI 2-sided [-4.3 to 0.3], Standard Error of Mean 1.39
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = -0.2, 90% CI 2-sided [-2.6 to 2.2], Standard Error of Mean 1.45
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 1.7, 90% CI 2-sided [-0.7 to 4.2], Standard Error of Mean 1.50
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = -1.2, 90% CI 2-sided [-3.6 to 1.2], Standard Error of Mean 1.45
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 0.1, 90% CI 2-sided [-2.4 to 2.6], Standard Error of Mean 1.51

24. Secondary Outcome: Percentage of Participants Achieving DLQI Total Score of 0 or 1 up to Week 16 - MR (FAS With Baseline >1, NRI)
Description: The Dermatology Life Quality Index (DLQI) is a general dermatology questionnaire that consists of 10 items that assess patient health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment) over the last week. Scoring for each item is on a qualitative 0 to 3 scale, with options of "Not at all", "A little", "A lot", "Very much". The scores are added up to a total composite score with the range from the minimum score of 0 to the maximum score of 30. The higher the score, the worse the outcomes. The assessments examined the percentage of patients with complete resolution of dermatology specific quality of life impact, as assessed by a total score of ≤ 1 (range: 0 - 30), where higher percentage indicates better improvement in DLQI.
Time Frame: At weeks 4, 8, 12 and 16
Population: All participants randomized and received at least one dose of study intervention with baseline >1 score were included.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 48 | 47 | 52 | 47
Percentage of Participants
  Week 4: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 4 | 6.8 [2.5 to 16.6] | 6.8 [2.5 to 16.6] | 8.9 [3.9 to 18.0] | 2.3 [0.2 to 9.4]
  Week 8: number analyzed (Participants) | 45 | 44 | 46 | 43
  Week 8 | 2.2 [0.2 to 9.2] | 6.8 [2.5 to 16.6] | 8.7 [3.8 to 17.6] | 4.7 [1.2 to 13.2]
  Week 12: number analyzed (Participants) | 45 | 44 | 46 | 43
  Week 12 | 4.4 [1.2 to 12.6] | 13.6 [6.1 to 24.3] | 10.9 [5.4 to 21.3] | 7.0 [2.6 to 17.0]
  Week 16: number analyzed (Participants) | 45 | 44 | 46 | 43
  Week 16 | 4.4 [1.2 to 12.6] | 4.5 [1.2 to 12.9] | 10.9 [5.4 to 21.3] | 11.6 [5.8 to 22.9]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 0.2, 90% CI 2-sided [-9.1 to 9.5], Standard Error of Mean 5.64
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 45mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = 1.2, 90% CI 2-sided [-7.4 to 9.8], Standard Error of Mean 5.25
Statistical Analysis 3: Comparison: Placebo vs PF-06826647 400mg QD; Week 4; Test type: Superiority; Risk Difference (RD) = -4.0, 90% CI 2-sided [-11.4 to 3.4], Standard Error of Mean 4.52
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = 4.3, 90% CI 2-sided [-3.3 to 11.8], Standard Error of Mean 4.57
Statistical Analysis 5: Comparison: Placebo vs PF-06700841 45mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = 6.2, 90% CI 2-sided [-1.8 to 14.2], Standard Error of Mean 4.87
Statistical Analysis 6: Comparison: Placebo vs PF-06826647 400mg QD; Week 8; Test type: Superiority; Risk Difference (RD) = 2.5, 90% CI 2-sided [-4.8 to 9.8], Standard Deviation 4.42
Statistical Analysis 7: Comparison: Placebo vs PF-06650833 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = 7.6, 90% CI 2-sided [-1.3 to 16.5], Standard Error of Mean 5.43
Statistical Analysis 8: Comparison: Placebo vs PF-06700841 45mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = 6.9, 90% CI 2-sided [-2.0 to 15.7], Standard Error of Mean 5.40
Statistical Analysis 9: Comparison: Placebo vs PF-06826647 400mg QD; Week 12; Test type: Superiority; Risk Difference (RD) = 2.9, 90% CI 2-sided [-5.5 to 11.3], Standard Error of Mean 5.09
Statistical Analysis 10: Comparison: Placebo vs PF-06650833 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 0.1, 90% CI 2-sided [-6.3 to 6.4], Standard Error of Mean 3.88
Statistical Analysis 11: Comparison: Placebo vs PF-06700841 45mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 6.5, 90% CI 2-sided [-2.8 to 15.7], Standard Error of Mean 5.63
Statistical Analysis 12: Comparison: Placebo vs PF-06826647 400mg QD; Week 16; Test type: Superiority; Risk Difference (RD) = 7.6, 90% CI 2-sided [-1.6 to 16.9], Standard Error of Mean 5.64

25. Secondary Outcome: Plasma Concentration Versus Time Summary (Pharmacokinetic Concentration Set)
Description: In summary statistics for pharmacokinetic, concentration values below the lower limit of quantification (LLOQ) was set to zero.
Time Frame: At weeks 1, 2, 4, 6, 8, 12 and 16
Population: All enrolled participants who took at least one dose of active PF-06700841, PF-06826647 or PF-06650833 and in whom at least one concentration value is reported.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/ml)
Arm/Group | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
Number analyzed (Participants) | 47 | 52 | 47
Nanograms per milliliter (ng/ml)
  WEEK 1 0H: number analyzed (Participants) | 35 | 41 | 31
  WEEK 1 0H | 31.79 (26.567) | 49.22 (64.871) | 281.7 (364.14)
  WEEK 2 0H: number analyzed (Participants) | 34 | 39 | 35
  WEEK 2 0H | 30.48 (35.796) | 51.48 (76.426) | 263.8 (388.42)
  WEEK 4 0H: number analyzed (Participants) | 39 | 41 | 32
  WEEK 4 0H | 25.33 (25.795) | 63.60 (77.180) | 215.6 (259.41)
  WEEK 6 0H: number analyzed (Participants) | 34 | 38 | 28
  WEEK 6 0H | 27.25 (29.905) | 47.38 (61.091) | 113.5 (140.62)
  WEEK 8 0H: number analyzed (Participants) | 35 | 43 | 31
  WEEK 8 0H | 34.72 (35.700) | 60.30 (92.758) | 277.2 (316.40)
  WEEK 8 30MIN: number analyzed (Participants) | 32 | 33 | 26
  WEEK 8 30MIN | 28.58 (24.510) | 254.7 (157.30) | 667.4 (560.37)
  WEEK 8 1H: number analyzed (Participants) | 32 | 35 | 28
  WEEK 8 1H | 45.70 (33.027) | 373.4 (174.51) | 817.2 (573.70)
  WEEK 8 2H: number analyzed (Participants) | 33 | 37 | 29
  WEEK 8 2H | 94.89 (48.222) | 296.0 (173.76) | 869.6 (549.58)
  WEEK 8 4H: number analyzed (Participants) | 34 | 38 | 30
  WEEK 8 4H | 112.4 (103.09) | 231.7 (168.11) | 784.8 (548.33)
  WEEK 12 0H: number analyzed (Participants) | 29 | 35 | 30
  WEEK 12 0H | 34.34 (32.046) | 52.95 (82.248) | 233.1 (322.19)
  WEEK 16 0H: number analyzed (Participants) | 24 | 32 | 25
  WEEK 16 0H | 39.41 (36.773) | 43.89 (67.413) | 244.4 (296.93)

ADVERSE EVENTS:
Time Frame: Up to 20 weeks.
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Placebo | PF-06650833 400mg QD | PF-06700841 45mg QD | PF-06826647 400mg QD
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47 | 0/52 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 2/47 | 0/52 | 2/47
Other Adverse Events (participants affected / at risk) | 6/48 | 10/47 | 14/52 | 18/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | PF-06650833 400mg QD (N=47) | PF-06700841 45mg QD (N=52) | PF-06826647 400mg QD (N=47)
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | PF-06650833 400mg QD (N=47) | PF-06700841 45mg QD (N=52) | PF-06826647 400mg QD (N=47)
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 3 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 4 | 6
Headache (Nervous system disorders) | 3 | 5 | 4 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 4 | 5 | 4
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT04092452/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT04092452/SAP_001.pdf